# Replication of the INSPIRE Trial in Healthcare Claims Data

# **DUPLICATE INSPIRE**

August 30, 2021

### 1. RCT Details

This section provides a high-level overview of an RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

### 1.1 Title

The Prevention of Chronic Obstructive Pulmonary Disease Exacerbations by Salmeterol/Fluticasone Propionate or Tiotropium Bromide (INSPIRE trial)

### 1.2 <u>Intended aim(s)</u>

The objective of the study is to compare the effect of the anti-inflammatory/bronchodilator combination of salmeterol/fluticasone propionate (SFC) with the bronchodilator tiotropium bromide on the rate of moderate and/or severe exacerbations during a 2-year treatment period, and secondarily on outcomes that might relate to exacerbations.

### 1.3 Primary endpoint for replication and RCT finding

Health care utilization exacerbation rate.

### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

With a sample size of 635 patients per treatment group, the trial will have 90% power to detect at least a 15% (equal to 1.445 exacerbations per subject per year) reduction in exacerbations in the SFC group at a two-sided significance level of alpha = 0.05

### 1.5 Trial estimate

Rate ratio = 0.967 (95% CI 0.836–1.119) comparing SFC to tiotropium bromide (Wedzicha et al., 2008, Am J Respir Crit Care Med). HR of 0.85 was used for power assessment based on RCT statistical analysis.

### 2. Person responsible for implementation of replication in Aetion

Helen Tesfaye, Pharm.D, ScM implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of design and analytic choices. All implementation steps are recorded, and implementation history is archived in the platform.

### 3. Data Source(s)

Optum Cliniformatics Data Mart, IBM MarketScan

### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expediated review

# Design Diagram - INSPIRE TRIAL REPLICATION



### 5. Cohort Identification

### 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score matched retrospective cohort study design comparing tiotropium to salmeterol. The patients will be required to have continuous enrollment during baseline period of 180 days before initiation of SFC or tiotropium inhalers (cohort entry date).

### 5.2 Important steps for cohort formation

New users (defined as no use in 180 days prior to index date) of an exposure and a comparator drug will be identified.

### 5.2.1 Eligible cohort entry date

SFC inhaler was first approved by FDA for market availability on August 24, 2000, and tiotropium on January 30, 2004

- Optum: January 30, 2004 March 31, 2020 (end of data availability is September 30, 2020 but excluded data generated during COVID-19 pandemic)
- Marketscan: January 30, 2004 December 31, 2018 (end of data availability)

### 5.2.2 Specify inclusion/exclusion criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

### 5.3 Flowchart of the study cohort assembly

| | OPTUM | | MARKETSCAN | |
|---|---|---|---|---|
| | Less Excluded | Remaining | Less Excluded | Remaining |
| | Patients | Patients | Patients | Patients |
| All patients | | 79,335,559 | | 200,203,908 |
| Did not meet cohort entry criteria | -77,381,938 | 1,953,621 | -196,683,354 | 3,520,554 |
| Excluded due to insufficient enrollment | -308,951 | 1,644,670 | -522,438 | 2,998,116 |
| Excluded due to prior use of referent | -274,142 | 1,370,528 | -362,567 | 2,635,549 |
| Excluded due to prior use of exposure | -641,980 | 728,548 | -1,225,388 | 1,410,161 |
| Excluded because patient qualified in >1 exposure category | -10,386 | 718,162 | -17,868 | 1,392,293 |

| Excluded based on Missing/Unknown Age | -6 | 718,156 | -1 | 1,392,292 |
|---|---|---|---|---|
| Excluded based on Missing/Unknown Gender | -125 | 718,031 | 0 | 1,392,292 |
| Excluded based on Inclusion #1 - Age 40 to 80 years old | -5 | 718,026 | 0 | 1,392,292 |
| Excluded based on Inclusion #3a - Diagnosis of COPD | -471,394 | 246,632 | -1,038,792 | 353,500 |
| Excluded based on Inclusion #3b - Clinical history of at least 1 COPD Exacerbation | -110,352 | 136,280 | -153,003 | 200,497 |
| Excluded based on Exclusion #1 - COPD exacerbation in the 6 weeks prior | -33,666 | 102,614 | -34,019 | 166,478 |
| Excluded based on Exclusion #2a - Current asthma | -13,344 | 89,270 | -13,539 | 152,939 |
| Excluded based on Exclusion #2b - Current eczema, atopic dermatitis and/or allergic rhinitis | -5,978 | 83,292 | -7,929 | 145,010 |
| Excluded based on Exclusion #3 - Has a known respiratory disorder other than COPD | -15,367 | 67,925 | -20,732 | 124,278 |
| Excluded based on Exclusion #4 - Has narrow-angle glaucoma, prostatic hyperplasia or | | | | |
| obstruction of the neck of the bladder | -3,927 | 63,998 | -5,648 | 118,630 |
| Excluded based on Exclusion #5 - Has undergone lung transplantation and/or lung volume | | | | |
| reduction | -11 | 63,987 | -41 | 118,589 |
| Excluded based on Exclusion #7 - Requires regular (daily) long-term oxygen therapy (LTOT) | -2,422 | 61,565 | -1,401 | 117,188 |
| Excluded based on Exclusion #8 - Is receiving beta-blockers (except eye drops) | -7,770 | 53,795 | -14,196 | 102,992 |
| Excluded based on Exclusion #11 - Has evidence of alcohol, drug or solvent abuse | -945 | 52,850 | -793 | 102,199 |
| Excluded based on Exclusion #14 - Exclude use of Salmeterol, tiotropium, and fluticasone | | | | |
| containing inhaler use | -591 | 52,259 | -819 | 101,380 |
| Final cohort | | 52,259 | | 101,380 |

### 6 Variables

### 6.1 Exposure-related variables:

### Study drug:

The study exposure of interest is initiation of SFC (LABA/ICS combination). Initiation will be defined by no use of inhaled SFC during the prior 180 days before treatment initiation (washout period).

### Comparator agents:

Initiators of tiotropium inhaler defined as no use of inhaled tiotropium during the 180 days prior to index date

Patients are required to be incident users with respect to both exposure groups.

### 6.2 Preliminary Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the default baseline covariate assessment period of 180 days prior to and including the index prescription date

Covariates listed above are a small subset of covariates that will ultimately be controlled in the design and analysis phase of the study. They are included in the preliminary assessment to determine the presence of adequate overlap between the two population of patients to proceed to the next phase of the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and initial power assessment and are listed in Table 1 (Appendix B).

### 6.3 Outcome variables and study follow-up:

### 6.3.1 Outcome variables

Effectiveness outcome variables of interest (definitions provided in **Appendix A**):

- Primary outcome: Healthcare utilization exacerbation rate per year (although the trial definition include 1) COPD hospitalizations or 2) exacerbations that required corticosteroids and/or antibiotics, in our emulation, we focused on 1) hospitalizations with COPD in the primary diagnosis position or 2) exacerbations that required corticosteroids. We did not include antibiotic use as part of the outcome definition because of our inability to determine whether the antibiotics were being used for COPD or some other indication)
- Secondary outcome:
  - All-cause death

Control outcomes of interest (control outcomes only serve to assess aspects of study validity but are not further interpreted): Pneumonia

### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analysis will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative rate of outcomes on treatment.

For the AT analysis, the follow-up will start the day after the initiation of SFC or tiotropium and will continue until the earliest date of the following events:

- The date of end of continued registration in the database,
- End of the study period or 730 days after cohort entry date,
- Death,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically
    provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this
    as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (SFC or tiotropium) + a 60-day grace period,
- The date of switching from an exposure to comparator and vice versa,
- The date of switching to or initiation of other LAMA (excluding tiotropium) and switch or initiation to other LABA/ICS (excluding SFC), LAMA/LABA, LABA only, LAMA/LABA/ICS combination, and ICS only inhalers.

For the ITT analyses, the censoring based on the switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

### 7 Initial Feasibility Analysis

Aetion report name:

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1742/rwrs/71660">https://bwh-dope.aetion.com/projects/details/1742/rwrs/71660</a>
Marketscan- <a href="https://bwh-dope.aetion.com/projects/details/1741/rwrs/71658">https://bwh-dope.aetion.com/projects/details/1741/rwrs/71658</a>

### Date conducted: 6/17/2021

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

### 8 Initial Power Assessment

### Aetion report name:

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1742/rwrs/71659">https://bwh-dope.aetion.com/projects/details/1742/rwrs/71659</a>
Marketscan- <a href="https://bwh-dope.aetion.com/projects/details/1741/rwrs/71657">https://bwh-dope.aetion.com/projects/details/1741/rwrs/71657</a>

### Date conducted: 6/17/2021

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index.

- Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.
- Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: |
|-------------------------|--------------|----------------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: |
| Reasons for stopping | | |
| analysis (if required): | | |

Effectiveness research with Real World Data to support FDA's regulatory decision making

### 9. Balance Assessment

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1742/rwrs/72363">https://bwh-dope.aetion.com/projects/details/1742/rwrs/72363</a>
Marketscan- <a href="https://bwh-dope.aetion.com/projects/details/1741/rwrs/72364">https://bwh-dope.aetion.com/projects/details/1741/rwrs/72364</a>

Date conducted: 7/14/2021

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

## • Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy outcome | 0 (0%) | 0 (0%) | 0 (0%) |
| Death | 706 (0.72%) | 368 (0.75%) | 338 (0.69%) |
| Start of an additional exposure | 8,037 (8.18%) | 4,562 (9.28%) | 3,475 (7.07%) |
| End of Index Exposure | 63,915 (65.03%) | 29,311 (59.65%) | 34,604 (70.42%) |
| Specified date reached | 2,286 (2.33%) | 1,069 (2.18%) | 1,217 (2.48%) |
| End of patient enrollment | 11,722 (11.93%) | 5,877 (11.96%) | 5,845 (11.89%) |
| Switch to other LABA, LAMA + LABA/LAMA combo + LAMA/LABA/ICS combo + ICS only + NH admissions Occurred | 11,612 (11.82%) | 7,952 (16.18%) | 3,660 (7.45%) |

### • Report follow-up time by treatment group.

| Patient Group | Optum<br>Median Follow-<br>Up Time (Days)<br>[IQR] | Marketscan<br>Median Follow-<br>Up Time (Days)<br>[IQR] |
|---|---|---|
| Overall Patient Population | 88 [88, 162] | 113 [88, 180] |
| Referent – Tiotropium | 88 [88, 160] | 99 [88, 175] |
| Exposure – Salmeterol/Fluticasone | 88 [88, 165] | 120 [88, 188] |

# • Report overall risk of the primary outcome.

| · | Optum | MarketScan | Pooled |
|-------------------------|--------|------------|--------|
| Risk per 1,000 patients | 152.99 | 138.80 | 143.63 |

### **10. Final Power Assessment**

Date conducted: 7/15/2021

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

| | ı |
|-------------------------------|-------------|
| Superiority Analysis (Pooled) | |
| Number of patients matched | |
| Reference | 49,138 |
| Exposed | 49,139 |
| Risk per 1,000 patients | 143.63 |
| Desired HR from RCT | 0.85 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 14115.52551 |
| Power | 1 |

| Superiority Analysis (Optum) | |
|------------------------------|-------------|
| Number of patients matched | |
| Reference | 18,017 |
| Exposed | 18,017 |
| Risk per 1,000 patients | 152.99 |
| Desired HR from RCT | 0.85 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 5512.84166 |
| Power | 0.999976837 |

| Superiority Analysis (Marketscan) | |
|-----------------------------------|------------|
| Number of patients matched | |
| Reference | 31,122 |
| Exposed | 31,122 |
| Risk per 1,000 patients | 138.80 |
| Desired HR from RCT | 0.85 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 8639.4672 |
| Power | 0.99999989 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: |
|-------------------------|--------------|----------------|
| Reviewed by FDA: | | Date reviewed: |
| Reasons for stopping | | |
| analysis (if required): | | |

### Appendix A: COPD Exacerbation (primary outcome), All-cause mortality (secondary outcome)

### **COPD Exacerbation**

Measured 1 day after drug initiation in primary diagnosis position specified below and inpatient care setting -

### **COPD** (Inpatient, Primary)

<u>ICD-9 Diagnosis</u>: 491.x, 492.x, 496 <u>ICD-10 Diagnosis</u>: J41.x, J42, J43.x, J44.x

### OR

Measured 1 day after drug initiation in any diagnosis position specified below and inpatient and outpatient care setting AND steroid use within 14 days -

### **COPD (Any care setting, Any position)**

<u>ICD-9 Diagnosis</u>: 491.x, 492.x, 496 ICD-10 Diagnosis: J41.x, J42, J43.x, J44.x

AND

### Corticosteroid systemic administration and/or oral prescription of --

- Prednisone
- Prednisolone
- Methylprednisolone
- Dexamethasone
- Hydrocortisone

\_\_\_\_\_

### **All-Cause Mortality**

Identified using the discharge status codes-

Optum-Inpatient/Outpatient

- 20 = EXPIRED
- 21 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 22 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 23 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 24 = EXPIRED TO BE DEFINED AT STATE LEVEL

- 25 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 26 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 27 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 28 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 29 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 40 = EXPIRED AT HOME (HOSPICE)
- 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE)
- 42 = EXPIRED PLACE UNKNOWN (HOSPICE)

### Marketscan-Inpatient

- 20 Died
- 22 Died
- 23 Died
- 24 Died
- 25 Died
- 26 Died
- 27 Died
- 28 Died
- 29 Died
- 40 Other died status or Expired at home (Hospice claims only) (depends on year)
- 41 Other died status or Expired in medical facility (Hospice claims only) (depends on year)
- 42 Other died status or Expired place unknown (Hospice claims only) (depends on year)
- 21 Died or Disch./Transf. to court/law enforcement (depends on year)

| # | INSPIRE trial definitions | Implementation in routine care | References/Rationale | Color coding |
|---|---|---|---|---|
| | | | Please see the following Google<br>drive for further details or any<br>missing information_<br>https://drive.google.com/drive/fold<br>ers/1WD618wrywYjEaXzfLTcuK- | |
| | Trial details-Intended S with label change - 2 weeks run-in | | VCcnb6b-gV | Criteria |
| | EXPOSURE vs. COMPARISON | | | Adequate mapping in claims |
| | Tiotropium 18 mcg once daily vs. Salmeterol/fluticasone propionate (SFC) 50/500 mcg twice daily | SFC vs. Tiotropium | | Intermediate mapping in |
| | Aim: To evaluate the effect of tiotropium compared to SFC on healthcare utilization of COPD exacerbations | Exposure: SFC Reference: Tiotropium | | claims |
| | PRIMARY OUTCOME | | | Poor mapping or cannot be measured in claims |
| | | Measured 1 day after drug initiation in primary diagnosis position and inpatient care setting | | |
| | Primary endpoint: Healthcare utilization COPD exacerbation rate | COPD (Inpatient, Primary) ICD-9 Diagnosis: 491.x, 492.x, 496 ICD-10 Diagnosis: J41.x, J42, J43.x, J44.x OR Measured 1 day after drug initiation in any diagnosis position any care setting AND steriod use within 14 days COPD (Any care setting, Any position) ICD-9 Diagnosis: 491.x, 492.x, 496 ICD-10 Diagnosis: J41.x, J42, J43.x, J44.x AND Corticosteriod systemic administration and/or oral prescription of: - Prednisone - Prednisolone - Methylprednisolone - Dexamethasone - Hydrocortisone | | Can't be measured in claims but not important for the analysis |
| | Tiotropium 18 mcg once daily vs. SFC 50/500 r | | | |
| | · | Age 40 to 80 years old at the time of drug initiation | | |
| 2 | Smoking history of ≥ 10 pack years | | | |
| 3a | Diagnosis of COPD | Measured from the start of all available data to and including the day of drug initiation in any diagnosis position and in the inpatient and outpatient care setting COPD ICD-9 Diagnosis: 491.x, 492.x, 496 ICD-10 Diagnosis: J41.x, J42, J43.x, J44.x | | |

| 3b | Clinical history of at least 1 COPD exacerbation | Measured since all available data to 43 days prior to drug initiation in primary diagnosis position and inpatient care setting COPD (Inpatient, Primary) ICD-9 Diagnosis: 491x, 492.x, 496.0 ICD-10 Diagnosis: J41, J42.x, J43.x, J44.x OR Measured since all available data to 43 days prior to drug initiation in any diagnosis position, inpatient and outpatient care setting AND steriod use within 30 days COPD ICD-9 Diagnosis: 491.x, 492.x, 496.0 ICD-10 Diagnosis: J41.x, J42, J43.x, J44.x AND Corticosteriod systemic administration and/or prescription - Prednisone - Prednisolone - Methylprednisolone - Methylprednisolone - Dexamethasone |
|---|---|---|
| 4 | Post bronchodilator FEV1 of < 50% of predicted normal | - Hydrocortisone |
| 5 | FEV1 / FVC ratio <70% | |
| 6 | Reversibility to 400 mcg albuterol of less or equal to 10% of predicted FEV1 at Visit 1 | |
| 7 | A score of 2 or more on the Modified Medical Research Council dyspnea scale | |
| 8 | Free from exacerbation in the 6 weeks prior to screening | Included in the exclusion criteria |
| | EXCLUSION CRITERIA | |
| 1 | COPD exacerbation in the 6 weeks prior to screening | Measured 42 days prior to and including the day of drug initiation in prescription claims COPD (Inpatient, Any) ICD-9 Diagnosis: 491.x, 492.x, 496.0 ICD-10 Diagnosis: J41.x, J42, J43.x, J44.x OR COPD (Any care setting, Any position) ICD-9 Diagnosis: 491.x, 492.x, 496.0 ICD-10 Diagnosis: J41.x, J42, J43.x, J44.x AND Corticosteriod systemic administration and/or prescription - Prednisone - Prednisolone - Methylprednisolone - Dexamethasone - Hydrocortisone |

| | | 7 |
|---|---|---|
| | | Measured 180 days prior to and including the day of drug initiation in any diagnosis position in the inpatient and outpatient care setting |
| | | A 11 /0 P: 111: 400 L 3 |
| | | Asthma (3 Diagnosis within 180 days) |
| | | ICD-9 Diagnosis: 493.x |
| | | ICD-10 Diagnosis: J45.x |
| | | <u>Eczema</u> |
| | | ICD-9 Diagnosis: 692.x |
| 2 | Current asthma, eczema, atopic dermatitis and/or allergic rhinitis | ICD-10 Diagnosis: L23.x, L24.x |
| | Current astrima, eczema, atopic dermatitis and/or anergic minitis | |
| | | Atopic dermatitis |
| | | ICD-9 Diagnosis: 691.x |
| | | ICD-10 Diagnosis: L20.x |
| | | To Diagnosis. E20.X |
| | | Allowed |
| | | Allergic rhinitis |
| I | | ICD-9 Diagnosis: 477.x |
| | | ICD10 Diagnosis: J30.x |
| <b>—</b> | | Measured since all available data to and including the day of drug initiation in any diagnosis |
| | | position in the inpatient and outpatient care setting |
| | | position in the imputions and outputions care setting |
| I | | Dulmanary Fibracia ay Interstitial Lung Disease (U.S.) |
| I | | Pulmonary Fibrosis or Interstitial Lung Disease (ILD) |
| | | ICD-9 Diagnosis: 515, 516.3x, 516.8, 516.9 |
| I | | ICD-10 Diagnosis: J84.10, J84.111, J84.112, J84.113, J84.114, J84.115, J84.116, J84.117, J84.09, |
| | | J84.2, J84.89, J84.9 |
| | | L |
| | | <u>Sarcoidosis</u> |
| | | ICD-9 diagnosis: 135 |
| | | ICD-10 diagnosis: D86.0, D86.2 |
| 3 | Has a known respiratory disorder other than COPD (e.g. lung cancer, sarcoidosis, tuberculosis or lung fibrosis) | <u>Lymphangioleiomyomatosis</u> |
| ľ | Thas a known respiratory disorder other than corp (e.g. rung cancer, sarcoldosis, tuberculosis or rung runosis) | ICD-9 diagnosis: 516.4 |
| | | ICD-10 diagnosis: J84.81 |
| | | Primary/Pulmonary Tuberculosis |
| | | ICD-9 diagnosis: 010.x, 011.x |
| | | ICD-10 diagnosis: A15.x |
| | | Cystic Fibrosis |
| I | | ICD-9 Diagnosis: 277.0x |
| | | ICD-10 Diagnosis: E84.xx |
| I | | Pulmonary Hypertension/Other Pulmonary Heart Disease |
| | | ICD-9 Diagnosis: 416 vy |
| | | Measured 180 days prior to and including the day of drug initiation in any diagnosis position in the inpatient and outpatient care setting |
| | | Narrow-angle Glaucoma |
| I | | |
| | | ICD-9 Diagnosis: 365.02, 36s.06, 365.2x |
| | | ICD-10 Diagnosis: H40.03x, H40.2xx, |
| | | Prostatic hyperplasia or obstruction of the neck of the bladder |
| I | Ulas paranu anala glaucama mastatia humanalasia ar abstruction of the mak of the hadder that in the continue of the | |
| 4 | Has narrow-angle glaucoma, prostatic hyperplasia or obstruction of the neck of the bladder that in the opinion of the | ICD-9 Diagnosis: 600.x |
| | investigator should prevent the subject from entering the study | ICD-10 Diagnosis: N40.x |
| | | OR |
| | | [ <del></del> |
| | | At least one 30-day supply presciption claims for oral: |
| | | Alfuzosin, doxazosin, tamsulosin, silodosin, finasteride 5 mg, dutasteride |

| _ | | Measured since all available data to and including the day of drug initiation in any diagnosis |
|---|---|---|
| | | position in the inpatient and outpatient care setting |
| | | Lung transplant |
| | | ICD-9 Diagnosis: V42.6, 996.84 |
| | | ICD-10 Diagnosis: Z94.2, T86.810, T86.811, T86.819 |
| | | ICD-9 Procedure: 33.5x ICD-10 Procedure: OBYMOZO, OBYMOZ1, OBYMOZ2, OBYKOZO, OBYKOZ1, OBYKOZ2, OBYLOZO, |
| | | OBYLOZ1, OBYLOZ2 |
| 5 | Has undergone lung transplantation and/or lung volume reduction | CPT-4 Code: 32850 - 32856 |
| | | Lung volume reduction surgery (LVRS) ICD-9 Procedure: 32.22, 32.3x |
| | | ICD-10 Procedure: 0BBC0ZZ, 0BBC4ZZ, 0BBD0ZZ, 0BBD4ZZ, 0BBF0ZZ, 0BBF4ZZ, 0BBG0ZZ, |
| | | OBBG4ZZ, OBBH0ZZ, OBBH4ZZ, OBBJ0ZZ, OBBJ4ZZ, OBBK0ZZ, OBBK4ZZ, OBBL0ZZ, OBBL4ZZ, |
| | | OBBMOZZ, OBBM4ZZ |
| | | CPT/HCPCS codes: 32491, 32672, G0302, G0303, G0304, G0305 |
| 6 | Female who is a nursing mother | |
| | | Measured since all available data to and including the day of drug initiation in any diagnosis |
| | | position in the inpatient and outpatient care setting |
| | | LTOT |
| 7 | Requires regular (daily) long-term oxygen therapy (LTOT) | ICD-9 Diagnosis: V46.2 |
| | | ICD-10 Diagnosis: Z99.81 |
| | | CPT/HCPCS code: E0424, E0441, E0443 |
| | | Measured 180 days prior to and including the day of drug initiation with prescription for oral: |
| | | Acebutolol, Atenolol, Betaxolol, Bisoprolol, Carteolol, Carvedilol, Labetalol, Metoprolol, |
| 8 | Is receiving beta-blockers (except eye drops) | Metiranolol, Nebivolol, Nadolol, Propranolol, Pindolol, Sotalol, Penbutolol, Oxprenolol |
| 9 | Has a serious, uncontrolled disease likely to interfere with the study | |
| 10 | Has received any other investigational drugs within the 4 weeks prior to Visit 1 | |
| | | Measured 180 days prior to and including the day of drug initiation in any diagnosis position in |
| | | the inpatient and outpatient care setting |
| | | Alcohol Abuse or Dependence |
| | | ICD-9 diagnosis: 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, |
| | | V11.3x |
| 11 | Has, in the opinion of the investigator, evidence of alcohol, drug or solvent abuse | ICD-10 diagnosis: F10.x, K70.x, G62.1, I42.6, 099.31x |
| | | Drug Abuse or Dependence |
| | | ICD-9 diagnosis: 292.xx, 304.xx, 305.2x-305.9x, 648.3x<br>ICD-10 diagnosis: F11.x, F12.x, F13.x, F14.x, F15.x, F16.x, F17.2x, F18.x, F19.x, F55.2, G62.0, |
| | | 099.32x |
| | | U99.32X |
| | | 099.52X |
| 12 | Has a known or suspected hypersensitivity to beta2-agonists, inhaled corticosteroids, anticholinergic agents or any components of the formulations (e.g. lactose or milk protein) | U99.32X |

| | | Measured 180 days prior to and including the day of drug initiation in prescription claims |
|---|---|---|
| 13 | Exclude use of Salmeterol, tiotropium, and fluticasone containing inhaler use within 180 days prior to CED | Brand names - STIOLTO RESPIMAT SEREVENT SEREVENT DISKUS ARNUITY ELLIPTA BREO ELLIPTA TRELEGY ELLIPTA FLOVENT HFA FLOVENT DISKUS ARMONAIR RESPICLICK ARMONAIR |
| | | OR Generic name - |
| | | TIOTROPIUM BROMIDE/OLODATEROL HCL<br>SALMETEROL XINAFOATE |

Optum MarketScan

### BEFORE PS MATCHING





The c-statistics for the propensity score model, pre-matching was 0.689. The post-matching c-statistic was 0.523.

The c-statistics for the propensity score model, pre-matching was 0.7. The post-matching c-statistic was 0.516.





### UNMATCHED

| UNIVIATCHED | | ODTUM | | | MADVETCCAN | | | POOLED | |
|---|---|---|---|---|---|---|---|---|---|
| | | OPTUM | | | MARKETSCAN | | | POOLED | |
| | Referent - Tiotropium | Exposure - Salmeterol/Fluticasone | St. Diff | Referent - Tiotropium | Exposure - Salmeterol/Fluticasone | St. Diff | Referent - Tiotropium | Exposure - Salmeterol/Fluticasone | St. Diff |
| Number of patients | 21,689 | 30,570 | | 36,727 | 64,653 | | 58,416 | 95,223 | |
| Calendar Time - Year of Initiation (2004 - 2020) | | | 0.4045 | | | 0.0100 | 6.070 (4.4.00) | 10.000 (10.00) | 0.010 |
| 2004-2006; n (%) | 1,330 (6.1%) | 3,505 (11.5%) | -0.1915 | 5,640 (15.4%) | 15,357 (23.8%) | -0.2128 | 6,970 (11.9%) | 18,862 (19.8%) | -0.218 |
| 2007-2008; n (%) | 2,190 (10.1%) | 3,669 (12.0%) | -0.0606 | 5,594 (15.2%) | 11,223 (17.4%) | -0.0596 | 7,784 (13.3%) | 14,892 (15.6%) | -0.065 |
| 2009-2011; n (%) | 4,060 (18.7%) | 6,299 (20.6%) | -0.0478 | 9,988 (27.2%) | 17,461 (27.0%) | 0.0045 | 14,048 (24.0%) | 23,760 (25.0%) | -0.023 |
| 2012-2015; n (%) | 6,704 (30.9%) | 8,124 (26.6%) | 0.0951 | 11,489 (31.3%) | 15,233 (23.6%) | 0.1732 | 18,193 (31.1%) | 23,357 (24.5%) | 0.148 |
| 2016-2018; n (%) | 5,091 (23.5%) | 6,116 (20.0%) | 0.0849 | 4,016 (10.9%) | 5,379 (8.3%) | 0.0883 | 9,107 (15.6%) | 11,495 (12.1%) | 0.101 |
| 2019-Mar. 2020; n (%) | 2,314 (10.7%) | 2,857 (9.3%) | 0.0467 | | | | 2,314 (10.7%) | 2,857 (9.3%) | 0.047 |
| DMG - Age | | | | | | | | | |
| mean (sd) | 67.67 (10.33) | 64.58 (13.34) | 0.2590 | 65.73 (11.22) | 62.49 (14.22) | 0.2530 | 66.45 (10.90) | 63.16 (13.94) | 0.263 |
| median [IQR] | 68.00 [60.00, 75.00] | 66.00 [56.00, 74.00] | 0.1676 | 64.00 [58.00, 74.00] | 62.00 [54.00, 73.00] | 0.1562 | 65.49 (10.90) | 63.28 (13.94) | 0.177 |
| DMG - Gender | | | | | | | , , | ì | |
| Male; n (%) | 7,779 (35.9%) | 10,307 (33.7%) | 0.0462 | 14,471 (39.4%) | 22,933 (35.5%) | 0.0806 | 22,250 (38.1%) | 33,240 (34.9%) | 0.067 |
| Female: n (%) | 13,910 (64.1%) | 20,263 (66.3%) | -0.0462 | 22,256 (60.6%) | 41.720 (64.5%) | -0.0806 | 36,166 (61.9%) | 61,983 (65.1%) | -0.067 |
| DMG - Geographic region | 15,510 (04.170) | 20,200 (00.070) | 0.0.02 | 22,230 (00.070) | 41,720 (04.570) | | 00,200 (02.07.2) | 52,000 (00.27.) | |
| Northeast; n (%) | 2,144 (9.9%) | 2,997 (9.8%) | 0.0034 | 5,662 (15.4%) | 10,090 (15.6%) | -0.0055 | 7,806 (13.4%) | 13,087 (13.7%) | -0.009 |
| South; n (%) | 9,881 (45.6%) | 13,979 (45.7%) | -0.0020 | 13,969 (38.0%) | 23,938 (37.0%) | 0.0207 | 23,850 (40.8%) | 37,917 (39.8%) | 0.020 |
| North Central; n (%) | 4.602 (21.2%) | 6.546 (21.4%) | -0.0049 | 12.524 (34.1%) | 21.068 (32.6%) | 0.0207 | 17,126 (29.3%) | 27,614 (29.0%) | 0.007 |
| West; n (%) | 5,062 (23.3%) | 7,048 (23.1%) | 0.0043 | 4,572 (12.4%) | 9,557 (14.8%) | -0.0701 | 9,634 (16.5%) | 16,605 (17.4%) | -0.024 |
| west; n (%) DRS - Combined comorbidity score, 180 days | 3,002 (23.3%) | 7,040 (23.170) | 0.0047 | 4,312 (12.4%) | 5,337 (14.0%) | 0.0701 | J,0J7 (10.J70) | 10,003 (17.470) | 0.024 |
| | 1.43 (1.73) | 1.20 (1.67) | 0.1353 | 1.13 (1.45) | 0.94 (1.39) | 0.1338 | 1.24 (1.56) | 1.02 (1.49) | 0.144 |
| mean (sd)median (IQR) | 1.43 (1.73) | 1.20 (1.67) | 0.0000 | 1.13 (1.45) | 1.00 [0.00, 1.00] | 0.0000 | 1.00 (1.56) | 1.02 (1.49) | 0.000 |
| median [ועא] DRS - Frailty Score: Empirical Version (mean) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.0000 | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 0.0000 | 1.00 (1.56) | 1.00 (1.49) | 0.000 |
| | 0.18 (0.06) | 0.17 (0.06) | 0.1667 | 0.17 (0.05) | 0.16 (0.05) | 0.2000 | 0.17 (0.05) | 0.16 (0.05) | 0.200 |
| mean (sd) | 0.18 (0.06) | 0.17 (0.06) | 0.1667 | 0.17 (0.05) | 0.15 [0.12, 0.18] | 0.2000 | 0.17 (0.05) | 0.15 (0.05) | 0.200 |
| median [IQR] | 0.17 [0.14, 0.21] | 0.16 [0.13, 0.20] | 0.1667 | 0.16 [0.13, 0.19] | 0.15 [0.12, 0.18] | 0.2000 | 0.16 (0.05) | 0.15 (0.05) | 0.200 |
| PLM-Smoking; n (%) | 6,731 (31.0%) | 5,954 (19.5%) | 0.2671 | 6,588 (17.9%) | 6,674 (10.3%) | 0.2197 | 13,319 (22.8%) | 12,628 (13.3%) | 0.249 |
| PLM-Pneumonia; n (%) | 1,409 (6.5%) | 1,750 (5.7%) | 0.0334 | 2,786 (7.6%) | 4,561 (7.1%) | 0.0192 | 4,195 (7.2%) | 6,311 (6.6%) | 0.024 |
| PLM - Oxygen usage; n (%) | 1,538 (7.1%) | 1,440 (4.7%) | 0.1020 | 3,158 (8.6%) | 3,635 (5.6%) | 0.1170 | 4,696 (8.0%) | 5,075 (5.3%) | 0.109 |
| PLM - Respiratory arrest/dependence on oxygen ; n (%) | 699 (3.2%) | 539 (1.8%) | 0.0898 | 1,088 (3.0%) | 1,177 (1.8%) | 0.0785 | 1,787 (3.1%) | 1,716 (1.8%) | 0.084 |
| PLM - CiPAP/BiPAP use; n (%) | 904 (4.2%) | 1,314 (4.3%) | -0.0050 | 1,943 (5.3%) | 3,038 (4.7%) | 0.0275 | 2,847 (4.9%) | 4,352 (4.6%) | 0.014 |
| PLM - Pulmonary rehabilitation ; n (%)* | 75 (0.3%) | 46 (0.2%) | 0.0200 | 150 (0.4%) | 103 (0.2%) | 0.0366 | 225 (0.4%) | 149 (0.2%) | 0.037 |
| PLM - Moderate COPD exacerbation - [Count with 365 to 181 days before CED]* | | | | | | | | | |
| mean (sd) | 1.37 (2.84) | 1.13 (2.47) | 0.0902 | 1.05 (2.25) | 0.83 (1.81) | 0.1077 | 1.17 (2.49) | 0.93 (2.05) | 0.105 |
| median [IQR] | 0.28 [0.00, 1.53] | 0.21 [0.00, 1.00] | 0.0263 | 0.05 [0.00, 1.00] | 0.08 [0.00, 1.00] | -0.0147 | 0.14 (2.49) | 0.12 (2.05) | 0.009 |
| PLM - Moderate COPD exacerbation - [Count 180 to 31 days before CED]* | | | | | | | | | |
| mean (sd) | 0.95 (2.07) | 0.72 (1.68) | 0.1220 | 0.68 (1.51) | 0.52 (1.22) | 0.1166 | 0.78 (1.74) | 0.58 (1.38) | 0.127 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.84] | 0.0000 | 0.00 [0.00, 0.81] | 0.00 [0.00, 0.66] | 0.0000 | 0.00 (1.74) | 0.00 (1.38) | 0.000 |
| PLM - Moderate COPD exacerbation - [Count with 30 days to CED]* | | | | | | | | | |
| mean (sd) | 0.02 (0.10) | 0.01 (0.08) | 0.1104 | 0.01 (0.08) | 0.01 (0.07) | 0.0000 | 0.01 (0.09) | 0.01 (0.07) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.09) | 0.00 (0.07) | 0.000 |
| PLM - Moderate exacerbations >=1 in 365 days before CED; n (%) | 15,357 (70.8%) | 21,008 (68.7%) | 0.0457 | 23,550 (64.1%) | 41,555 (64.3%) | -0.0042 | 38,907 (66.6%) | 62,563 (65.7%) | 0.019 |
| PLM - Moderate exacerbations >= 2 in 365 days before CED ; n (%) | 9,947 (45.9%) | 11,428 (37.4%) | 0.1731 | 13,956 (38.0%) | 19,175 (29.7%) | 0.1761 | 23,903 (40.9%) | 30,603 (32.1%) | 0.184 |
| PLM - Severe COPD exacerbation - [Count with 365 to 181 days before CED] * | | | | | | | | | |
| mean (sd) | 0.03 (0.18) | 0.03 (0.17) | 0.0000 | 0.05 (0.21) | 0.04 (0.19) | 0.0499 | 0.04 (0.20) | 0.04 (0.18) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.20) | 0.00 (0.18) | 0.000 |
| PLM - Severe COPD exacerbation - [Count with 180 to 31 days before CED] * | | | | | | | | | |
| mean (sd) | 0.02 (0.14) | 0.02 (0.12) | 0.0000 | 0.03 (0.16) | 0.02 (0.14) | 0.0665 | 0.03 (0.15) | 0.02 (0.13) | 0.071 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.15) | 0.00 (0.13) | 0.000 |
| PLM - Severe COPD exacerbation - [Count with 30 days lookback] * | | | | | | | | | |
| mean (sd) | 0.00 (0.01) | 0.00 (0.01) | 0.0000 | 0.00 (0.01) | 0.00 (0.01) | 0.0000 | 0.00 (0.01) | 0.00 (0.01) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.01) | 0.00 (0.01) | 0.000 |
| PLM - Severe exacerbations >=1 in 365 days before CED; n (%) | 1,333 (6.1%) | 1,499 (4.9%) | 0.0527 | 3,221 (8.8%) | 4,394 (6.8%) | 0.0746 | 4,554 (7.8%) | 5,893 (6.2%) | 0.063 |
| PLM - Severe exacerbations >=2 in 365 days before CED; n (%) | 118 (0.5%) | 128 (0.4%) | 0.0149 | 265 (0.7%) | 326 (0.5%) | 0.0259 | 383 (0.7%) | 454 (0.5%) | 0.026 |
| PLM - GOLD C/D Status ; n (%) | 7,067 (32.6%) | 7,801 (25.5%) | 0.1569 | 12,368 (33.7%) | 16,852 (26.1%) | 0.1666 | 19,435 (33.3%) | 24,653 (25.9%) | 0.163 |
| PRX - LABA only; n (%) | 299 (1.4%) | 100 (0.3%) | 0.1200 | 1,170 (3.2%) | 338 (0.5%) | 0.2014 | 1,469 (2.5%) | 438 (0.5%) | 0.165 |
| PRX - LAMA (except tiotropium) inhalers ; n (%) | 123 (0.6%) | 159 (0.5%) | 0.0135 | 184 (0.5%) | 175 (0.3%) | 0.0317 | 307 (0.5%) | 334 (0.4%) | 0.015 |
| PRX - ICS only inhalers ; n (%) | 2,727 (12.6%) | 4,010 (13.1%) | -0.0149 | 6,319 (17.2%) | 11,104 (17.2%) | 0.0000 | 9,046 (15.5%) | 15,114 (15.9%) | -0.011 |
| PRX - LABA/LAMA inhaler use ; n (%) | 146 (0.7%) | 96 (0.3%) | 0.0567 | 83 (0.2%) | 45 (0.1%) | 0.0258 | 229 (0.4%) | 141 (0.1%) | 0.060 |
| PRX - Other LABA/ICS combination ; n (%) | 3,473 (16.0%) | 901 (2.9%) | 0.4595 | 5,501 (15.0%) | 1,484 (2.3%) | 0.4638 | 8,974 (15.4%) | 2,385 (2.5%) | 0.464 |
| PRX - COPD Maintenance therapy inhalers ; n (%) | 3,942 (18.2%) | 1,224 (4.0%) | 0.4640 | 6,296 (17.1%) | 1,719 (2.7%) | 0.4968 | 10,238 (17.5%) | 2,943 (3.1%) | 0.488 |
| PRX - SAMA inhaler use ; n (%) | 765 (3.5%) | 1,171 (3.8%) | -0.0160 | 1,653 (4.5%) | 2,912 (4.5%) | 0.0000 | 2,418 (4.1%) | 4,083 (4.3%) | -0.010 |
| PRX - SABA use ; n (%) | 10,165 (46.9%) | 14,075 (46.0%) | 0.0180 | 16,966 (46.2%) | 29,037 (44.9%) | 0.0261 | 27,131 (46.4%) | 43,112 (45.3%) | 0.022 |
| PRX - SABA/SAMA use; n (%) | 2,485 (11.5%) | 3,905 (12.8%) | -0.0398 | 4,865 (13.2%) | 9,933 (15.4%) | -0.0629 | 7,350 (12.6%) | 13,838 (14.5%) | -0.056 |
| PRX - Antibiotics treatment (180 days to 31 days before CED); n (%) | 8,080 (37.3%) | 11,493 (37.6%) | -0.0062 | 14,869 (40.5%) | 27,269 (42.2%) | -0.0345 | 22,949 (39.3%) | 38,762 (40.7%) | -0.029 |
| | | | _ | | | | | | |

| BBV 4 - 111 - 1 | 2 225 (1.1.20) | 5 070 (40 000) | 0.4345 | 6.046 (47.00) | 11.051 (00.00) | -0.1504 | 0.242/45.00() | 20 722 (24 00() | 0.440 |
|---|---|---|---|---|---|---|---|---|---|
| PRX - Antibiotics treatment (30 days to CED); n (%) | 3,096 (14.3%)<br>6,911 (31.9%) | 5,872 (19.2%) | -0.1315<br>-0.0107 | 6,246 (17.0%) | 14,851 (23.0%)<br>20.935 (32.4%) | -0.1504 | 9,342 (16.0%)<br>18,504 (31.7%) | 20,723 (21.8%)<br>30,848 (32.4%) | -0.149<br>-0.015 |
| PRX - Systemic Corticosteroids (with CPT) (180 days to 31 days before CED); n (%) PRX - Systemic Corticosteroids (with CPT) (30 days to CED); n (%) | 1,106 (5.1%) | 9,913 (32.4%)<br>3,126 (10.2%) | -0.0107 | 11,593 (31.6%)<br>2,576 (7.0%) | 8,168 (12.6%) | -0.0172 | 3,682 (6.3%) | 11,294 (11.9%) | -0.015 |
| PRX - Systemic Controsteroids (With CPT) (50 days to CED); II (%) | 67 (0.3%) | 42 (0.1%) | 0.0448 | 162 (0.4%) | 76 (0.1%) | 0.0601 | 229 (0.4%) | 118 (0.1%) | 0.060 |
| PRX - ROHUHHIASE, II (%) | 67 (0.3%) | 42 (0.1%) | 0.0448 | 182 (0.4%) | 76 (0.1%) | 0.0001 | 223 (0.470) | 110 (0.174) | 0.000 |
| CVD - Unstable angina/MI; n (%) | 593 (2.7%) | 643 (2.1%) | 0.0392 | 701 (1.9%) | 1,029 (1.6%) | 0.0229 | 1,294 (2.2%) | 1,672 (1.8%) | 0.029 |
| CVD - Stable Angina ; n (%) | 403 (1.9%) | 486 (1.6%) | 0.0229 | 573 (1.6%) | 834 (1.3%) | 0.0251 | 976 (1.7%) | 1,320 (1.4%) | 0.024 |
| CVD - Any Heart failure (HF); n (%) | 1,334 (6.2%) | 1,649 (5.4%) | 0.0342 | 2,076 (5.7%) | 3,132 (4.8%) | 0.0404 | 3,410 (5.8%) | 4,781 (5.0%) | 0.035 |
| CVD - Atrial fibrillation; n (%) | 1,091 (5.0%) | 1,261 (4.1%) | 0.0432 | 1,764 (4.8%) | 2,458 (3.8%) | 0.0493 | 2,855 (4.9%) | 3,719 (3.9%) | 0.049 |
| CVD - Other dysrythmias ; n (%)* | 1,576 (7.3%) | 1,894 (6.2%) | 0.0439 | 2,195 (6.0%) | 3,210 (5.0%) | 0.0439 | 3,771 (6.5%) | 5,104 (5.4%) | 0.047 |
| CVD - Valve disorder ; n (%) | 277 (1.3%) | 332 (1.1%) | 0.0184 | 336 (0.9%) | 612 (0.9%) | 0.0000 | 613 (1.0%) | 944 (1.0%) | 0.000 |
| CVD - Implantable cardioverter defibrillator ; n (%)* | 69 (0.3%) | 82 (0.3%) | 0.0000 | 111 (0.3%) | 109 (0.2%) | 0.0200 | 180 (0.3%) | 191 (0.2%) | 0.020 |
| CVD - CABG/PCI; n (%) | 521 (2.4%) | 534 (1.7%) | 0.0494 | 464 (1.3%) | 595 (0.9%) | 0.0384 | 985 (1.7%) | 1,129 (1.2%) | 0.042 |
| CVD - Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 2,581 (11.9%) | 2,968 (9.7%) | 0.0709 | 4,121 (11.2%) | 5,577 (8.6%) | 0.0871 | 6,702 (11.5%) | 8,545 (9.0%) | 0.082 |
| CVD - Stroke/TIA ; n (%) | 641 (3.0%) | 713 (2.3%) | 0.0436 | 943 (2.6%) | 1,546 (2.4%) | 0.0128 | 1,584 (2.7%) | 2,259 (2.4%) | 0.019 |
| CVD - Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) | 1,693 (7.8%) | 1,661 (5.4%) | 0.0968 | 1,776 (4.8%) | 2,384 (3.7%) | 0.0545 | 3,469 (5.9%) | 4,045 (4.2%) | 0.078 |
| CVD - Hyperlipidemia ; n (%) | 9,573 (44.1%) | 12,176 (39.8%) | 0.0872 | 10,218 (27.8%) | 15,419 (23.8%) | 0.0915 | 19,791 (33.9%) | 27,595 (29.0%) | 0.106 |
| CVD - Hypertension; n (%) | 11,323 (52.2%) | 14,593 (47.7%) | 0.0901 | 13,871 (37.8%) | 21,783 (33.7%) | 0.0856 | 25,194 (43.1%) | 36,376 (38.2%) | 0.100 |
| CRX - ACEi or ARB; n (%) | 8,168 (37.7%) | 11,243 (36.8%) | 0.0186 | 13,292 (36.2%) | 22,744 (35.2%) | 0.0209 | 21,460 (36.7%) | 33,987 (35.7%) | 0.021 |
| CRX - Mineralocorticoid receptor antagonist ; n (%) | 325 (1.5%) | 516 (1.7%) | -0.0159 | 778 (2.1%) | 1,227 (1.9%) | 0.0143 | 1,103 (1.9%) | 1,743 (1.8%) | 0.007 |
| CRX - Loop or Thiazide diuretics; n (%) | 4,670 (21.5%) | 6,398 (20.9%) | 0.0147 | 8,382 (22.8%) | 14,759 (22.8%) | 0.0000 | 13,052 (22.3%) | 21,157 (22.2%) | 0.002 |
| CRX - Statins and other lipid lowering agents; n (%) | 8,977 (41.4%) | 11,512 (37.7%) | 0.0757 | 14,474 (39.4%) | 23,089 (35.7%) | 0.0765 | 23,451 (40.1%) | 34,601 (36.3%) | 0.078 |
| CRX - CCB and other antihypertensives; n (%) | 4,813 (22.2%) | 6,332 (20.7%) | 0.0365 | 8,069 (22.0%) | 13,275 (20.5%) | 0.0367 | 12,882 (22.1%) | 19,607 (20.6%) | 0.037 |
| CRX - Digoxin ; n (%)* | 314 (1.4%) | 440 (1.4%) | 0.0000 | 923 (2.5%) | 1,584 (2.5%) | 0.0000 | 1,237 (2.1%) | 2,024 (2.1%) | 0.000 |
| CRX - Nitrates; n (%)* | 702 (3.2%) | 908 (3.0%) | 0.0115 | 1,615 (4.4%) | 2,613 (4.0%) | 0.0199 | 2,317 (4.0%) | 3,521 (3.7%) | 0.016 |
| OCM - Type 1 or 2 DM; n (%) | 4,453 (20.5%) | 6,394 (20.9%) | -0.0099 | 6,166 (16.8%) | 10,874 (16.8%) | 0.0000 | 10,619 (18.2%) | 17,268 (18.1%) | 0.003 |
| OCM - Occurrence of Diabetic retinopathy/nephropathy/neuropathy; n (%)* | 1,266 (5.8%) | 1,801 (5.9%) | -0.0043 | 1,080 (2.9%) | 1,727 (2.7%) | 0.0121 | 2,346 (4.0%) | 3,528 (3.7%) | 0.016 |
| OCM - Hypertensive nephropathy; n (%)* | 689 (3.2%) | 848 (2.8%) | 0.0235 | 453 (1.2%) | 611 (0.9%) | 0.0294 | 1,142 (2.0%) | 1,459 (1.5%) | 0.010 |
| OCM-Hypotension ; n (%)* | 383 (1.8%) | 423 (1.4%) | 0.0319 | 466 (1.3%) | 621 (1.0%) | 0.0281 | 849 (1.5%) | 1,044 (1.1%) | 0.035 |
| OCM - Hyperkalemia ; n (%)* | 210 (1.0%) | 269 (0.9%) | 0.0103 | 219 (0.6%) | 297 (0.5%) | 0.0135 | 429 (0.7%) | 566 (0.6%) | 0.012 |
| OCM - CKD II, III, or IV; n (%) | 1,196 (5.5%) | 1,533 (5.0%) | 0.0224 | 665 (1.8%) | 968 (1.5%) | 0.0236 | 1,861 (3.2%) | 2,501 (2.6%) | 0.036 |
| OCM - HD/PD/ESRD; n (%)* | 73 (0.3%) | 96 (0.3%) | 0.0000 | 155 (0.4%) | 268 (0.4%) | 0.0000 | 228 (0.4%) | 364 (0.4%) | 0.000 |
| OCM - Osteoporosis; n (%) | 2,569 (11.8%) | 3,180 (10.4%) | 0.0446 | 3,643 (9.9%) | 5,889 (9.1%) | 0.0273 | 6,212 (10.6%) | 9,069 (9.5%) | 0.037 |
| OCM - Sleep apnea ; n (%) | 2,011 (9.3%) | 2,533 (8.3%) | 0.0353 | 3,369 (9.2%) | 4,832 (7.5%) | 0.0615 | 5,380 (9.2%) | 7,365 (7.7%) | 0.054 |
| OCM-Fractures ; n (%) | 939 (4.3%) | 1,250 (4.1%) | 0.0100 | 1,631 (4.4%) | 2,887 (4.5%) | -0.0048 | 2,570 (4.4%) | 4,137 (4.3%) | 0.005 |
| OCM - Other Arthritis, Arthropathies and Musculoskeletal Pain ; n (%) | 7,847 (36.2%) | 11,143 (36.5%) | -0.0062 | 11,173 (30.4%) | 20,027 (31.0%) | -0.0130 | 19,020 (32.6%) | 31,170 (32.7%) | -0.002 |
| OCM - Dorsopathies; n (%) | 6,114 (28.2%) | 8,136 (26.6%) | 0.0359 | 8,276 (22.5%) | 13,884 (21.5%) | 0.0241 | 14,390 (24.6%) | 22,020 (23.1%) | 0.035 |
| OCM - Gout (acute/chronic) ; n (%)* | 143 (0.7%) | 251 (0.8%) | -0.0116 | 278 (0.8%) | 437 (0.7%) | 0.0116 | 421 (0.7%) | 688 (0.7%) | 0.000 |
| OCM - Hyperthyroidism ; n (%)* | 136 (0.6%) | 171 (0.6%) | 0.0000 | 179 (0.5%) | 286 (0.4%) | 0.0149 | 315 (0.5%) | 457 (0.5%) | 0.000 |
| OCM - Hypothyroidism ; n (%)* | 2,033 (9.4%) | 2,899 (9.5%) | -0.0034 | 2,650 (7.2%) | 4,532 (7.0%) | 0.0078 | 4,683 (8.0%) | 7,431 (7.8%) | 0.007 |
| OCM - VTE; n (%)* | 400 (1.8%) | 502 (1.6%) | 0.0155 | 663 (1.8%) | 1,090 (1.7%) | 0.0076 | 1,063 (1.8%) | 1,592 (1.7%) | 0.008 |
| OCM - GERD ; n (%) | 3,134 (14.4%) | 3,995 (13.1%) | 0.0378 | 2,891 (7.9%) | 4,522 (7.0%) | 0.0343 | 6,025 (10.3%) | 8,517 (8.9%) | 0.048 |
| OCM-Cancer; n (%) | 2,248 (10.4%) | 2,942 (9.6%) | 0.0267 | 3,071 (8.4%) | 4,758 (7.4%) | 0.0371 | 5,319 (9.1%) | 7,700 (8.1%) | 0.036 |
| OCM - Hypovolemia/volume depletion ; n (%)* | 468 (2.2%) | 601 (2.0%) | 0.0139 | 622 (1.7%) | 1,021 (1.6%) | 0.0079 | 1,090 (1.9%) | 1,622 (1.7%) | 0.015 |
| OCM-Anemia ; n (%) | 2,185 (10.1%) | 3,009 (9.8%) | 0.0100 | 2,840 (7.7%) | 4,754 (7.4%) | 0.0114 | 5,025 (8.6%) | 7,763 (8.2%) | 0.014 |
| OCM - Dementia ; n (%)* | 777 (3.6%) | 968 (3.2%) | 0.0221 | 887 (2.4%) | 1,320 (2.0%) | 0.0273 | 1,664 (2.8%) | 2,288 (2.4%) | 0.025 |
| OCM - Depression ; n (%) | 3,467 (16.0%) | 4,284 (14.0%) | 0.0560 | 3,580 (9.7%) | 5,735 (8.9%) | 0.0275 | 7,047 (12.1%) | 10,019 (10.5%) | 0.051 |
| SOUL ALL COLONIA COLON | 2 222 (42 42) | 0.400/40.40/ | 0.0000 | 0.404/0.50/ | E 075 (0 40() | 0.0242 | F 224 (0 40/) | 0.057.0.500 | 0.041 |
| ORX - Metformin; n (%)* | 2,200 (10.1%) | 3,182 (10.4%) | -0.0099 | 3,134 (8.5%) | 5,875 (9.1%) | -0.0212 | 5,334 (9.1%) | 9,057 (9.5%) | -0.014 |
| ORX - 1st and 2nd Generation SUs ; n (%) ORX - Insulins : n (%) | 1,054 (4.9%)<br>897 (4.1%) | 1,597 (5.2%) | -0.0137<br>-0.0149 | 1,837 (5.0%) | 3,494 (5.4%)<br>2.879 (4.5%) | -0.0180<br>-0.0147 | 2,891 (4.9%)<br>2,448 (4.2%) | 5,091 (5.3%)<br>4,234 (4.4%) | -0.018<br>-0.010 |
| ORX - Insulins ; n (%) ORX - Other antidiabetic medications use; n (%) | 897 (4.1%)<br>826 (3.8%) | 1,355 (4.4%)<br>1,179 (3.9%) | -0.0149 | 1,551 (4.2%)<br>1,704 (4.6%) | 2,879 (4.5%)<br>3.252 (5.0%) | -0.0147 | 2,530 (4.3%) | 4,234 (4.4%) | -0.010 |
| | 5,118 (23.6%) | 1,179 (3.9%)<br>6,819 (22.3%) | 0.0309 | | 3,252 (5.0%)<br>13,897 (21.5%) | -0.0187 | 12,953 (22.2%) | 20,716 (21.8%) | 0.019 |
| ORX - PPIs or H2RAs use; n (%)* ORX - NSAIDs ; n (%)* | 5,118 (23.6%)<br>3,492 (16.1%) | 5,242 (17.1%) | -0.0269 | 7,835 (21.3%)<br>6,115 (16.6%) | 13,897 (21.5%) | -0.0500 | 9,607 (16.4%) | 17,189 (18.1%) | -0.045 |
| ORX - NSAIDS; n (%)* ORX - Use of opioids; n (%)* | 7,529 (34.7%) | 10,709 (35.0%) | -0.0269 | 13,564 (36.9%) | 23,859 (36.9%) | 0.0000 | 21,093 (36.1%) | 34,568 (36.3%) | -0.045 |
| ORX - Use of antipsychotics ; n (%)* | 992 (4.6%) | 1,281 (4.2%) | 0.0195 | 1,445 (3.9%) | 2,380 (3.7%) | 0.0105 | 2,437 (4.2%) | 3,661 (3.8%) | 0.020 |
| ORX - Use of antidepressants : n (%) | 7,865 (36.3%) | 10,356 (33.9%) | 0.0503 | 12,794 (34.8%) | 21,535 (33.3%) | 0.0103 | 20,659 (35.4%) | 31,891 (33.5%) | 0.040 |
| ORX - Use of anxiolytics/hypnotics; n (%) | 2,098 (9.7%) | 3,001 (9.8%) | -0.0034 | 3,956 (10.8%) | 7,101 (11.0%) | -0.0064 | 6,054 (10.4%) | 10,102 (10.6%) | -0.007 |
| ORX - Use of anticonvulsants ; n (%)* | 3,680 (17.0%) | 4,802 (15.7%) | 0.0352 | 4,975 (13.5%) | 8,461 (13.1%) | 0.0118 | 8,655 (14.8%) | 13,263 (13.9%) | 0.026 |
| ORX - Use of Benzodiazepines ; n (%)* | 3,637 (16.8%) | 5,129 (16.8%) | 0.0000 | 8,276 (22.5%) | 13,795 (21.3%) | 0.0290 | 11,913 (20.4%) | 18,924 (19.9%) | 0.012 |
| ORX - Use of dementia meds ; n (%)* | 546 (2.5%) | 679 (2.2%) | 0.0198 | 871 (2.4%) | 1,357 (2.1%) | 0.0202 | 1,417 (2.4%) | 2,036 (2.1%) | 0.020 |
| ORX - Use of antiparkinsonian meds ; n (%)* | 821 (3.8%) | 997 (3.3%) | 0.0270 | 1,231 (3.4%) | 2,000 (3.1%) | 0.0169 | 2,052 (3.5%) | 2,997 (3.1%) | 0.022 |
| ORX - Use of oral anticoagulants ; n (%)* | 1,035 (4.8%) | 1,345 (4.4%) | 0.0191 | 2,074 (5.6%) | 3,252 (5.0%) | 0.0268 | 3,109 (5.3%) | 4,597 (4.8%) | 0.023 |
| ORX - Use of antiplatelet agents ; n (%)* | 1,438 (6.6%) | 1,582 (5.2%) | 0.0594 | 3,661 (10.0%) | 5,416 (8.4%) | 0.0554 | 5,099 (8.7%) | 6,998 (7.3%) | 0.052 |
| | · · · · · | | | | | | | | |
| LFS - Obesity; n (%) | 1,630 (7.5%) | 2,388 (7.8%) | -0.0113 | 1,578 (4.3%) | 2,791 (4.3%) | 0.0000 | 3,208 (5.5%) | 5,179 (5.4%) | 0.004 |
| PFT - Spirometry test only; n (%) | 4,594 (21.2%) | 3,785 (12.4%) | 0.2370 | 9,392 (25.6%) | 10,035 (15.5%) | 0.2519 | 13,986 (23.9%) | 13,820 (14.5%) | 0.240 |
| PFT - Spirometry test only (Count - 180 days to 31 days before CED) * | | | | | | | | | |
| mean (sd) | 0.22 (0.74) | 0.13 (0.55) | 0.1380 | 0.23 (0.70) | 0.15 (0.53) | 0.1289 | 0.23 (0.72) | 0.14 (0.54) | 0.141 |

| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.72) | 0.00 (0.54) | 0.000 |
|---|---|---|---|---|---|---|---|---|---|
| PFT - Spirometry test only (Count - 30 days to CED) * | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.72) | 0.00 (0.54) | 0.000 |
| mean (sd) | 0.18 (0.62) | 0.08 (0.41) | 0.1903 | 0.20 (0.60) | 0.09 (0.39) | 0.2174 | 0.19 (0.61) | 0.09 (0.40) | 0.194 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.61) | 0.00 (0.40) | 0.000 |
| PFT - Lung volume, Diffuse capacity, pulmonary stress testing (any); n (%) | 2,852 (13.1%) | 2,795 (9.1%) | 0.1276 | 4,207 (11.5%) | 5,282 (8.2%) | 0.1109 | 7,059 (12.1%) | 8,077 (8.5%) | 0.119 |
| Title Eding volume, Dinase capacity, pullionally seriess reseming (any), it (70) | 2,032 (13.170) | 2,755 (5.176) | 0.1270 | 4,207 (11.576) | 3,202 (0.270) | 0.1103 | 7,033 (12.170) | 0,017 (0.370) | 0.113 |
| HCU - Pulmonologist visit (180 to 1 day before CED); n (%) | 290 (1.3%) | 246 (0.8%) | 0.0491 | 7,544 (20.5%) | 8,804 (13.6%) | 0.1843 | 7,834 (13.4%) | 9,050 (9.5%) | 0.123 |
| HCU - Pulmonologist visit on CED; n (%) | 43 (0.2%) | 28 (0.1%) | 0.0258 | 1,568 (4.3%) | 1,216 (1.9%) | 0.1388 | 1,611 (2.8%) | 1,244 (1.3%) | 0.106 |
| HCU - Pulmonologist visit (Number of during CAP) * | | , , | | | | | | | |
| mean (sd) | 0.08 (1.11) | 0.05 (0.93) | 0.0293 | 0.89 (2.39) | 0.49 (1.77) | 0.1902 | 0.59 (2.01) | 0.35 (1.55) | 0.134 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (2.01) | 0.00 (1.55) | 0.000 |
| HCU - Number of Internal Medicine/Family Medicine Visits | | | | | | | | | |
| mean (sd) | 7.62 (11.28) | 6.95 (11.33) | 0.0593 | 6.26 (10.74) | 5.66 (9.03) | 0.0605 | 6.76 (10.94) | 6.07 (9.83) | 0.066 |
| median [IQR] | 4.00 [1.00, 10.00] | 3.00 [0.00, 9.00] | 0.0885 | 4.00 [1.00, 8.00] | 3.00 [1.00, 7.00] | 0.1008 | 4.00 (10.94) | 3.00 (9.83) | 0.096 |
| HCU - Number of Cardiologist visits | | | | | | | | | |
| mean (sd) | 0.89 (3.16) | 0.75 (2.76) | 0.0472 | 0.81 (2.83) | 0.67 (2.84) | 0.0494 | 0.84 (2.96) | 0.70 (2.81) | 0.049 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (2.96) | 0.00 (2.81) | 0.000 |
| HCU - Number of Emergency Department (ED) visits v3 | | | | | | | | | |
| mean (sd) | 0.47 (1.31) | 0.42 (1.18) | 0.0401 | 0.17 (1.10) | 0.16 (1.10) | 0.0091 | 0.28 (1.18) | 0.24 (1.13) | 0.035 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (1.18) | 0.00 (1.13) | 0.000 |
| HCU - Old hospitalization (-180 days to -31 days before CED); n (%) | 1,883 (8.7%) | 2,196 (7.2%) | 0.0555 | 4,861 (13.2%) | 7,875 (12.2%) | 0.0300 | 6,744 (11.5%) | 10,071 (10.6%) | 0.029 |
| HCU - Recent hospitalization (-30 days to CED date); n (%) | 202 (0.9%) | 264 (0.9%) | 0.0000 | 595 (1.6%) | 1,252 (1.9%) | -0.0229 | 797 (1.4%) | 1,516 (1.6%) | -0.016 |
| HCU - Number of hospitalizations during CAP | | | | | | | | | |
| mean (sd) | 0.11 (0.38) | 0.09 (0.35) | 0.0547 | 0.16 (0.43) | 0.16 (0.43) | 0.0000 | 0.14 (0.41) | 0.14 (0.41) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.41) | 0.00 (0.41) | 0.000 |
| HCU - Blood eosinophilia or Serum IgE test order; n (%)* | 109 (0.5%) | 161 (0.5%) | 0.0000 | 145 (0.4%) | 299 (0.5%) | -0.0149 | 254 (0.4%) | 460 (0.5%) | -0.015 |
| HCU - Pneumococcal vaccine; n (%) | 2,791 (12.9%) | 3,065 (10.0%) | 0.0912 | 2,119 (5.8%) | 2,509 (3.9%) | 0.0885 | 4,910 (8.4%) | 5,574 (5.9%) | 0.097 |
| HCU - Flu vaccine ; n (%) | 4,134 (19.1%) | 5,214 (17.1%) | 0.0520 | 4,507 (12.3%) | 6,971 (10.8%) | 0.0469 | 8,641 (14.8%) | 12,185 (12.8%) | 0.058 |
| HCU - Bone mineral density ; n (%) | 988 (4.6%) | 1,210 (4.0%) | 0.0296 | 1,146 (3.1%) | 1,659 (2.6%) | 0.0301 | 2,134 (3.7%) | 2,869 (3.0%) | 0.039 |
| HCU - Pap smear ; n (%) | 817 (3.8%) | 1,594 (5.2%) | -0.0676 | 1,625 (4.4%) | 4,095 (6.3%) | -0.0845 | 2,442 (4.2%) | 5,689 (6.0%) | -0.082 |
| HCU - Mammogram ; n (%) | 2,744 (12.7%) | 3,954 (12.9%) | -0.0060 | 3,874 (10.5%) | 7,572 (11.7%) | -0.0382 | 6,618 (11.3%) | 11,526 (12.1%) | -0.025 |
| HCU - Prostate exam for DRE; n (%) | 694 (3.2%) | 751 (2.5%) | 0.0421 | 666 (1.8%) | 767 (1.2%) | 0.0494 | 1,360 (2.3%) | 1,518 (1.6%) | 0.051 |
| HCU - Number of Echocardiogram * | | | | | | | | | |
| mean (sd) | 0.20 (1.26) | 0.17 (1.13) | 0.0251 | 0.22 (0.79) | 0.21 (0.80) | 0.0126 | 0.21 (0.99) | 0.20 (0.92) | 0.010 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.99) | 0.00 (0.92) | 0.000 |
| HCU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) | 992 (4.6%) | 1,258 (4.1%) | 0.0245 | 1,950 (5.3%) | 3,230 (5.0%) | 0.0136 | 2,942 (5.0%) | 4,488 (4.7%) | 0.014 |
| HCU - Number of Distinct Medication Prescriptions (not generalized to generics) | | | | | | | | | |
| mean (sd) | 20.64 (17.20) | 20.20 (16.75) | 0.0259 | 19.54 (14.98) | 19.61 (15.46) | -0.0046 | 19.95 (15.84) | 19.80 (15.89) | 0.009 |
| median [IQR] | 16.00 [9.00, 27.00] | 16.00 [9.00, 27.00] | 0.0000 | 16.00 [9.00, 26.00] | 16.00 [9.00, 26.00] | 0.0000 | 16.00 (15.84) | 16.00 (15.89) | 0.000 |
| SES - Copay for pharmacy cost (charges in U.S. \$) | | | 0.0246 | | | 0.0057 | 20 42 (24 20) | 20 42 (20 05) | 0.000 |
| mean (sd) | 32.20 (38.19) | 33.47 (36.20) | -0.0341 | 26.20 (26.21) | 26.05 (26.49) | 0.0057 | 28.43 (31.20) | 28.43 (29.95) | 0.000 |
| median [IQR] | 23.64 [9.89, 41.20] | 25.69 [12.25, 43.02] | -0.0551 | 20.87 [10.38, 35.00] | 21.04 [10.00, 35.00] | -0.0065 | 21.90 (31.20) | 22.53 (29.95) | -0.021 |
| SES - Business type | | | 0.2525 | | | + | | | 0.252 |
| Commercial; n (%) | 6,697 (30.9%) | 13,136 (43.0%) | -0.2527 | | 1 | | 6,697 (30.9%) | 13,136 (43.0%) | -0.253 |
| Medicare; n (%) | 14,992 (69.1%) | 17,434 (57.0%) | 0.2527 | | | + | 14,992 (69.1%) | 17,434 (57.0%) | 0.253 |
| SES - Low income indicator ; n (%) | 4,586 (21.1%) | 4,970 (16.3%) | 0.1233 | | 1 | | 4,586 (21.1%) | 4,970 (16.3%) | 0.123 |
| SES - Insurance Plan type | | | + | 10.555 (00.00) | 15 00 1 /0 5 01/ | 0.0070 | 40.050/00.00/ | 10.001/00.00 | 0.05= |
| Comprehensive; n (%) | | | + | 10,656 (29.0%) | 16,804 (26.0%) | 0.0672 | 10,656 (29.0%) | 16,804 (26.0%) | 0.067 |
| HMO; n (%) | | ļ | 1 | 4,376 (11.9%) | 8,310 (12.9%) | -0.0303 | 4,376 (11.9%) | 8,310 (12.9%) | -0.030 |
| PPO; n (%) | | ļ | 1 | 17,092 (46.5%) | 30,849 (47.7%) | -0.0240 | 17,092 (46.5%) | 30,849 (47.7%) | -0.024 |
| Others; n (%) | | l . | | 4,603 (12.5%) | 8,690 (13.4%) | -0.0268 | 4,603 (12.5%) | 8,690 (13.4%) | -0.027 |

<sup>\*</sup> Not included in PS model

| PS MATCHED | OPTUM | | | - | MARKETSCAN | POOLED | | | |
|---|---|---|---|---|---|---|---|---|---|
| Number of patients | Referent - Tiotropium<br>18,017 | Exposure - Salmeterol/Fluticasone<br>18,017 | St. Diff | Referent - Tiotropium<br>31,122 | Exposure - Salmeterol/Fluticasone<br>31,122 | St. Diff | Referent - Tiotropium<br>49,139 | Exposure - Salmeterol/Fluticasone<br>49,139 | e St. Diff |
| Calendar Time - Year of Initiation (2004 - 2020) | 18,017 | 18,017 | | 31,122 | 31,122 | | 49,139 | 49,139 | + |
| 2004-2006; n (%) | 1,289 (7.2%) | 1,219 (6.8%) | 0.0157 | 5,326 (17.1%) | 5,292 (17.0%) | 0.0027 | 6,615 (13.5%) | 6,511 (13.3%) | 0.006 |
| 2007-2008; n (%) | 2,030 (11.3%) | 2,065 (11.5%) | -0.0063 | 5,203 (16.7%) | 5,279 (17.0%) | -0.0080 | 7,233 (14.7%) | 7,344 (14.9%) | -0.006 |
| 2009-2011; n (%) | 3,594 (19.9%) | 3,602 (20.0%) | -0.0025 | 8,529 (27.4%) | 8,599 (27.6%) | -0.0045 | 12,123 (24.7%) | 12,201 (24.8%) | -0.002 |
| 2012-2015; n (%) | 5,440 (30.2%) | 5,414 (30.0%) | 0.0044 | 9,009 (28.9%) | 8,912 (28.6%) | 0.0066 | 14,449 (29.4%) | 14,326 (29.2%) | 0.004 |
| 2016-2018; n (%) | 3,880 (21.5%) | 3,887 (21.6%) | -0.0024 | 3,055 (9.8%) | 3,040 (9.8%) | 0.0000 | 6,935 (14.1%) | 6,927 (14.1%) | 0.000 |
| 2019-Mar. 2020; n (%) | 1,784 (9.9%) | 1,830 (10.2%) | -0.0100 | | | | 1,784 (9.9%) | 1,830 (10.2%) | -0.010 |
| DMG - Age | | | | | | | | | + |
| mean (sd) | 67.43 (10.50) | 67.84 (11.57) | -0.0371 | 65.64 (11.34) | 66.01 (12.78) | -0.0306 | 66.30 (11.04) | 66.68 (12.35) | -0.032 |
| median [IQR] | 68.00 [60.00, 75.00] | 69.00 [60.00, 76.00] | -0.0905 | 64.00 [58.00, 74.00] | 65.00 [57.00, 76.00] | -0.0828 | 65.47 (11.04) | 66.47 (12.35) | -0.085 |
| DMG - Gender | | | | | | | 10.000 (00.00) | | |
| Male; n (%) | 6,330 (35.1%) | 6,304 (35.0%) | 0.0021 | 12,025 (38.6%) | 12,000 (38.6%) | 0.0000 | 18,355 (37.4%) | 18,304 (37.2%) | 0.004 |
| Female; n (%) DMG - Geographic region | 11,687 (64.9%) | 11,713 (65.0%) | -0.0021 | 19,097 (61.4%) | 19,122 (61.4%) | 0.0000 | 30,784 (62.6%) | 30,835 (62.8%) | -0.004 |
| Northeast: n (%) | 1,731 (9.6%) | 1,705 (9.5%) | 0.0034 | 4,713 (15.1%) | 4,752 (15.3%) | -0.0056 | 6,444 (13.1%) | 6,457 (13.1%) | 0.000 |
| South; n (%) | 8,144 (45.2%) | 8,102 (45.0%) | 0.0040 | 11,758 (37.8%) | 11,766 (37.8%) | 0.0000 | 19,902 (40.5%) | 19,868 (40.4%) | 0.002 |
| North Central; n (%) | 3,811 (21.2%) | 3,855 (21.4%) | -0.0049 | 10,606 (34.1%) | 10,593 (34.0%) | 0.0021 | 14,417 (29.3%) | 14,448 (29.4%) | -0.002 |
| West; n (%) | 4,331 (24.0%) | 4,355 (24.2%) | -0.0047 | 4,045 (13.0%) | 4,011 (12.9%) | 0.0030 | 8,376 (17.0%) | 8,366 (17.0%) | 0.000 |
| DRS - Combined comorbidity score, 180 days | | | | | | | | | 1 |
| mean (sd) | 1.37 (1.71) | 1.38 (1.78) | -0.0057 | 1.10 (1.45) | 1.10 (1.52) | 0.0000 | 1.20 (1.55) | 1.20 (1.62) | 0.000 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.0000 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.0000 | 1.00 (1.55) | 1.00 (1.62) | 0.000 |
| DRS - Frailty Score: Empirical Version (mean) | | | | | | | | 2 4 7 (2 2 2) | |
| mean (sd) | 0.18 (0.06) | 0.18 (0.06) | 0.0000 | 0.17 (0.05) | 0.17 (0.06) | 0.0000 | 0.17 (0.05) | 0.17 (0.06) | 0.000 |
| median [IQR] | 0.17 [0.14, 0.21] | 0.17 [0.14, 0.21] | 0.0000 | 0.16 [0.13, 0.19] | 0.15 [0.13, 0.19] | 0.1811 | 0.16 (0.05) | 0.16 (0.06) | 0.000 |
| PLM - Smoking ; n (%) | 4,968 (27.6%) | 4,844 (26.9%) | 0.0157 | 4,977 (16.0%) | 4,803 (15.4%) | 0.0165 | 9,945 (20.2%) | 9,647 (19.6%) | 0.015 |
| PLM - Pneumonia ; n (%) | 1,122 (6.2%) | 1,104 (6.1%) | 0.0042 | 2,335 (7.5%) | 2,288 (7.4%) | 0.0038 | 3,457 (7.0%) | 3,392 (6.9%) | 0.004 |
| PLM - Oxygen usage; n (%) | 1,135 (6.3%) | 1,127 (6.3%) | 0.0000 | 2,474 (7.9%) | 2,436 (7.8%) | 0.0037 | 3,609 (7.3%) | 3,563 (7.3%) | 0.000 |
| PLM - Respiratory arrest/dependence on oxygen ; n (%) | 452 (2.5%) | 452 (2.5%) | 0.0000 | 791 (2.5%) | 735 (2.4%) | 0.0065 | 1,243 (2.5%) | 1,187 (2.4%) | 0.006 |
| PLM - CiPAP/BiPAP use; n (%) | 706 (3.9%) | 715 (4.0%) | -0.0051 | 1,569 (5.0%) | 1,544 (5.0%) | 0.0000 | 2,275 (4.6%) | 2,259 (4.6%) | 0.000 |
| PLM - Pulmonary rehabilitation ; n (%)* | 49 (0.3%) | 36 (0.2%) | 0.0200 | 99 (0.3%) | 78 (0.3%) | 0.0000 | 148 (0.3%) | 114 (0.2%) | 0.020 |
| PLM - Moderate COPD exacerbation - [Count with 365 to 181 days before CED]* | | | | | | | | | |
| mean (sd) | 1.27 (2.69) | 1.30 (2.75) | -0.0110 | 0.98 (2.17) | 0.97 (2.04) | 0.0047 | 1.09 (2.37) | 1.09 (2.33) | 0.000 |
| median [IQR] | 0.22 [0.00, 1.35] | 0.27 [0.00, 1.40] | -0.0184 | 0.01 [0.00, 1.00] | 0.05 [0.00, 1.00] | -0.0190 | 0.09 (2.37) | 0.13 (2.33) | -0.017 |
| PLM - Moderate COPD exacerbation - [Count 180 to 31 days before CED]*mean (sd) | 0.86 (1.93) | 0.82 (1.84) | 0.0212 | 0.63 (1.44) | 0.62 (1.42) | 0.0070 | 0.71 (1.64) | 0.69 (1.59) | 0.012 |
| median (su) | 0.00 [0.00, 0.95] | 0.00 [0.00, 0.93] | 0.0000 | 0.00 [0.00, 0.75] | 0.00 [0.00, 0.75] | 0.0000 | 0.00 (1.64) | 0.00 (1.59) | 0.000 |
| PLM - Moderate COPD exacerbation - [Count with 30 days to CED]* | 0.00 [0.00, 0.93] | 0.00 [0.00, 0.93] | 0.0000 | 0.00 [0.00, 0.73] | 0.00 [0.00, 0.73] | 0.0000 | 0.00 (1.04) | 0.00 (1.55) | 0.000 |
| mean (sd) | 0.02 (0.10) | 0.01(0.09) | 0.1051 | 0.01 (0.08) | 0.01 (0.08) | 0.0000 | 0.01 (0.09) | 0.01 (0.08) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.09) | 0.00 (0.08) | 0.000 |
| PLM - Moderate exacerbations >=1 in 365 days before CED; n (%) | 12,493 (69.3%) | 12,555 (69.7%) | -0.0087 | 19,559 (62.8%) | 19,638 (63.1%) | -0.0062 | 32,052 (65.2%) | 32,193 (65.5%) | -0.006 |
| PLM - Moderate exacerbations >= 2 in 365 days before CED; n (%) | 7,747 (43.0%) | 7,755 (43.0%) | 0.0000 | 11,085 (35.6%) | 11,239 (36.1%) | -0.0104 | 18,832 (38.3%) | 18,994 (38.7%) | -0.008 |
| PLM - Severe COPD exacerbation - [Count with 365 to 181 days before CED] * | | | | | | | | | |
| mean (sd) | 0.03 (0.18) | 0.03 (0.18) | 0.0000 | 0.05 (0.21) | 0.05 (0.21) | 0.0000 | 0.04 (0.20) | 0.04 (0.20) | 0.000 |
| median [IQR] PLM - Severe COPD exacerbation - [Count with 180 to 31 days before CED] * | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.20) | 0.00 (0.20) | 0.000 |
| PLM - Severe COPD exacerbation - [Count with 180 to 31 days before CED] *mean (sd) | 0.02 (0.14) | 0.02 (0.13) | 0.0000 | 0.03 (0.15) | 0.03 (0.15) | 0.0000 | 0.03 (0.15) | 0.03 (0.14) | 0.000 |
| median (Su) | 0.02 (0.14) | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.15) | 0.00 (0.14) | 0.000 |
| PLM - Severe COPD exacerbation - [Count with 30 days lookback] * | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 3.0000 | 0.00 (0.13) | 0.00 (0.1-1) | + 0.000 |
| mean (sd) | 0.00 (0.01) | 0.00 (0.01) | 0.0000 | 0.00 (0.01) | 0.00 (0.01) | 0.0000 | 0.00 (0.01) | 0.00 (0.01) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.01) | 0.00 (0.01) | 0.000 |
| PLM - Severe exacerbations >=1 in 365 days before CED; n (%) | 1,038 (5.8%) | 1,015 (5.6%) | 0.0086 | 2,595 (8.3%) | 2,650 (8.5%) | -0.0072 | 3,633 (7.4%) | 3,665 (7.5%) | -0.004 |
| PLM - Severe exacerbations >=2 in 365 days before CED ; n (%) | 93 (0.5%) | 86 (0.5%) | 0.0000 | 198 (0.6%) | 198 (0.6%) | 0.0000 | 291 (0.6%) | 284 (0.6%) | 0.000 |
| PLM - GOLD C/D Status ; n (%) | 5,385 (29.9%) | 5,395 (29.9%) | 0.0000 | 9,771 (31.4%) | 9,873 (31.7%) | -0.0065 | 15,156 (30.8%) | 15,268 (31.1%) | -0.006 |
| PRX - LABA only ; n (%) | 93 (0.5%) | 99 (0.5%) | 0.0000 | 348 (1.1%) | 332 (1.1%) | 0.0000 | 441 (0.9%) | 431 (0.9%) | 0.000 |
| PRX - LAMA (except tiotropium) inhalers; n (%) | 79 (0.4%) | 129 (0.7%) | -0.0406 | 104 (0.3%) | 160 (0.5%) | -0.0317 | 183 (0.4%) | 289 (0.6%) | -0.028 |
| PRX - ICS only inhalers; n (%) | 2,225 (12.3%) | 2,173 (12.1%) | 0.0061 | 5,212 (16.7%) | 5,163 (16.6%) | 0.0027 | 7,437 (15.1%) | 7,336 (14.9%) | 0.006 |
| PRX - LABA/LAMA inhaler use ; n (%) | 114 (0.6%) | 80 (0.4%) | 0.0284 | 56 (0.2%) | 42 (0.1%) | 0.0258 | 170 (0.3%) | 122 (0.2%) | 0.020 |
| PRX - Other LABA/ICS combination ; n (%) | 916 (5.1%) | 892 (5.0%) | 0.0046 | 1,495 (4.8%) | 1,469 (4.7%) | 0.0047 | 2,411 (4.9%) | 2,361 (4.8%) | 0.005 |
| PRX - COPD Maintenance therapy inhalers; n (%) | 1,183 (6.6%) | 1,169 (6.5%) | 0.0040 | 1,729 (5.6%) | 1,698 (5.5%) | 0.0044 | 2,912 (5.9%) | 2,867 (5.8%) | 0.004 |
| PRX - SAMA inhaler use; n (%) | 656 (3.6%) | 654 (3.6%) | 0.0000 | 1,405 (4.5%) | 1,431 (4.6%) | -0.0048 | 2,061 (4.2%) | 2,085 (4.2%) | 0.000 |
| PRX - SABA use; n (%) | 8,121 (45.1%) | 8,083 (44.9%) | 0.0040 | 13,827 (44.4%) | 13,671 (43.9%) | 0.0101 | 21,948 (44.7%) | 21,754 (44.3%) | 0.008 |
| PRX - SABA/SAMA use; n (%) | 2,035 (11.3%) | 2,140 (11.9%) | -0.0187 | 4,133 (13.3%) | 4,220 (13.6%) | -0.0088 | 6,168 (12.6%) | 6,360 (12.9%) | -0.009 |
| PRX - Antibiotics treatment (180 days to 31 days before CED); n (%) | 6,629 (36.8%) | 6,636 (36.8%) | 0.0000 | 12,467 (40.1%) | 12,337 (39.6%) | 0.0102 | 19,096 (38.9%) | 18,973 (38.6%) | 0.006 |
| PRX - Antibiotics treatment (30 days to CED); n (%) | 2,690 (14.9%) | 2,627 (14.6%) | 0.0085 | 5,514 (17.7%) | 5,441 (17.5%) | 0.0053 | 8,204 (16.7%) | 8,068 (16.4%) | 0.008 |
| PRX - Systemic Corticosteroids (with CPT) use (180 to 31 days before CED); n (%) | 5,612 (31.1%) | 5,577 (31.0%) | 0.0022 | 9,580 (30.8%) | 9,597 (30.8%) | 0.0000 | 15,192 (30.9%) | 15,174 (30.9%) | 0.000 |

| PRX - Systemic Corticosteroids (with CPT) use (30 days to CED); n (%) | 1,016 (5.6%) | 940 (5.2%) | 0.0177 | 2,352 (7.6%) | 2,284 (7.3%) | 0.0114 | 3,368 (6.9%) | 3,224 (6.6%) | 0.012 |
|---|---|---|---|---|---|---|---|---|---|
| PRX - Roflumilast; n (%) * | 40 (0.2%) | 31 (0.2%) | 0.0000 | 102 (0.3%) | 53 (0.2%) | 0.0200 | 142 (0.3%) | 084 (0.2%) | 0.020 |
| CMB. Hastald and the 160 | 450 (2.59() | 464 (2.69) | 0.0000 | FOC (4.00() | 500 (4.00/) | 0.0000 | 1,064 (2.2%) | 1,062 (2.2%) | 0.000 |
| CVD - Unstable angina/MI; n (%) CVD - Stable Angina : n (%) | 468 (2.6%)<br>318 (1.8%) | 464 (2.6%)<br>314 (1.7%) | 0.0000 | 596 (1.9%)<br>482 (1.5%) | 598 (1.9%)<br>476 (1.5%) | 0.0000 | 800 (1.6%) | 790 (1.6%) | 0.000 |
| CVD - Any Heart failure (HF); n (%) | 1,108 (6.1%) | 1,131 (6.3%) | -0.0083 | 1,797 (5.8%) | 1,807 (5.8%) | 0.0000 | 2,905 (5.9%) | 2,938 (6.0%) | -0.004 |
| CVD - Atrial fibrillation; n (%) | 911 (5.1%) | 911 (5.1%) | 0.0000 | 1,480 (4.8%) | 1,488 (4.8%) | 0.0000 | 2,391 (4.9%) | 2,399 (4.9%) | 0.000 |
| CVD - Other dysrythmias ; n (%)* | 1,256 (7.0%) | 1,324 (7.3%) | -0.0116 | 1,788 (5.7%) | 1,841 (5.9%) | -0.0086 | 3,044 (6.2%) | 3,165 (6.4%) | -0.008 |
| CVD - Valve disorder ; n (%) | 231 (1.3%) | 232 (1.3%) | 0.0000 | 289 (0.9%) | 283 (0.9%) | 0.0000 | 520 (1.1%) | 515 (1.0%) | 0.010 |
| CVD - Implantable cardioverter defibrillator ; n (%)* | 51 (0.3%) | 59 (0.3%) | 0.0000 | 94 (0.3%) | 67 (0.2%) | 0.0200 | 145 (0.3%) | 126 (0.3%) | 0.000 |
| CVD - CABG/PCI; n (%) | 407 (2.3%) | 400 (2.2%) | 0.0067 | 375 (1.2%) | 359 (1.2%) | 0.0000 | 782 (1.6%) | 759 (1.5%) | 0.008 |
| CVD - Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 2,082 (11.6%) | 2,082 (11.6%) | 0.0000 | 3,397 (10.9%) | 3,423 (11.0%) | -0.0032 | 5,479 (11.2%) | 5,505 (11.2%) | 0.000 |
| CVD - Stroke/TIA ; n (%) | 512 (2.8%) | 525 (2.9%) | -0.0060<br>0.0000 | 808 (2.6%) | 814 (2.6%) | 0.0000<br>0.0047 | 1,320 (2.7%)<br>2,815 (5.7%) | 1,339 (2.7%)<br>2,808 (5.7%) | 0.000 |
| CVD - Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) CVD - Hyperlipidemia; n (%) | 1,333 (7.4%)<br>7.804 (43.3%) | 1,330 (7.4%)<br>7,866 (43.7%) | -0.0081 | 1,482 (4.8%)<br>8.374 (26.9%) | 1,478 (4.7%)<br>8,401 (27.0%) | -0.0023 | 16,178 (32.9%) | 16,267 (33.1%) | -0.004 |
| CVD - Hypertension; n (%) | 9,269 (51.4%) | 9,370 (52.0%) | -0.0120 | 11,614 (37.3%) | 11,709 (37.6%) | -0.0062 | 20,883 (42.5%) | 21,079 (42.9%) | -0.008 |
| CTO TYPE CENSOR, TO (A) | 3,203 (31.470) | 3,370 (32.070) | | 11,014 (37.370) | 11,703 (37.070) | 0.000 | 20,000 (12,07.) | ==,0.00(1=1011) | |
| CRX - ACEi or ARB; n (%) | 6,749 (37.5%) | 6,860 (38.1%) | -0.0124 | 11,265 (36.2%) | 11,481 (36.9%) | -0.0145 | 18,014 (36.7%) | 18,341 (37.3%) | -0.012 |
| CRX - Mineralocorticoid receptor antagonist ; n (%) | 268 (1.5%) | 300 (1.7%) | -0.0159 | 654 (2.1%) | 655 (2.1%) | 0.0000 | 922 (1.9%) | 955 (1.9%) | 0.000 |
| CRX - Loop or Thiazide diuretics; n (%) | 3,888 (21.6%) | 3,980 (22.1%) | -0.0121 | 7,188 (23.1%) | 7,276 (23.4%) | -0.0071 | 11,076 (22.5%) | 11,256 (22.9%) | -0.010 |
| CRX - Statins and other lipid lowering agents; n (%) | 7,327 (40.7%) | 7,417 (41.2%) | -0.0102 | 12,165 (39.1%) | 12,317 (39.6%) | -0.0102 | 19,492 (39.7%) | 19,734 (40.2%) | -0.010 |
| CRX - CCB and other antihypertensives; n (%) | 3,956 (22.0%) | 4,018 (22.3%) | -0.0072 | 6,868 (22.1%) | 6,911 (22.2%) | -0.0024 | 10,824 (22.0%) | 10,929 (22.2%) | -0.005 |
| CRX - Digoxin ; n (%)* CRX - Nitrates: n (%)* | 279 (1.5%)<br>585 (3.2%) | 299 (1.7%)<br>585 (3.2%) | -0.0159<br>0.0000 | 804 (2.6%)<br>1,392 (4.5%) | 874 (2.8%)<br>1,445 (4.6%) | -0.0123<br>-0.0048 | 1,083 (2.2%)<br>1,977 (4.0%) | 1,173 (2.4%)<br>2,030 (4.1%) | -0.013<br>-0.005 |
| CRA - NILI ates; II (%) | 585 (3.2%) | 585 (5.2%) | 0.0000 | 1,392 (4.5%) | 1,445 (4.6%) | -0.0048 | 1,977 (4.0%) | 2,030 (4.1%) | -0.005 |
| OCM - Type 1 or 2 DM; n (%) | 3,731 (20.7%) | 3,818 (21.2%) | -0.0123 | 5,268 (16.9%) | 5,288 (17.0%) | -0.0027 | 8,999 (18.3%) | 9,106 (18.5%) | -0.005 |
| OCM - Occurrence of Diabetic retinopathy/nephropathy/neuropathy; n (%)* | 1,023 (5.7%) | 1,174 (6.5%) | -0.0334 | 914 (2.9%) | 942 (3.0%) | -0.0059 | 1,937 (3.9%) | 2,116 (4.3%) | -0.020 |
| OCM - Hypertensive nephropathy; n (%)* | 557 (3.1%) | 600 (3.3%) | -0.0114 | 379 (1.2%) | 377 (1.2%) | 0.0000 | 936 (1.9%) | 977 (2.0%) | -0.007 |
| OCM-Hypotension; n (%)* | 300 (1.7%) | 292 (1.6%) | 0.0079 | 389 (1.2%) | 353 (1.1%) | 0.0094 | 689 (1.4%) | 645 (1.3%) | 0.009 |
| OCM - Hyperkalemia ; n (%)* | 170 (0.9%) | 191 (1.1%) | -0.0201 | 185 (0.6%) | 170 (0.5%) | 0.0135 | 355 (0.7%) | 361 (0.7%) | 0.000 |
| OCM-CKD II, III, or IV; n (%) | 994 (5.5%) | 1,011 (5.6%) | -0.0044 | 565 (1.8%) | 578 (1.9%) | -0.0074 | 1,559 (3.2%) | 1,589 (3.2%) | 0.000 |
| OCM-HD/PD/ESRD; n (%)* | 60 (0.3%) | 63 (0.3%) | 0.0000 | 129 (0.4%) | 161 (0.5%) | -0.0149 | 189 (0.4%) | 224 (0.5%) | -0.015 |
| OCM - Osteoporosis; n (%) | 2,105 (11.7%)<br>1.533 (8.5%) | 2,099 (11.7%) | 0.0000 | 3,085 (9.9%) | 3,127 (10.0%) | -0.0033<br>0.0036 | 5,190 (10.6%)<br>4,172 (8.5%) | 5,226 (10.6%)<br>4,122 (8.4%) | 0.000 |
| OCM - Sleep apnea ; n (%) OCM - Fractures : n (%) | 1,533 (8.5%)<br>792 (4.4%) | 1,510 (8.4%)<br>795 (4.4%) | 0.0000 | 2,639 (8.5%)<br>1,410 (4.5%) | 2,612 (8.4%)<br>1,453 (4.7%) | -0.0036 | 4,172 (8.5%)<br>2,202 (4.5%) | 4,122 (8.4%)<br>2,248 (4.6%) | -0.005 |
| OCM - Practures ; n (%) OCM - Other Arthritis, Arthropathies and Musculoskeletal Pain ; n (%) | 6.547 (36.3%) | 6.597 (36.6%) | -0.0062 | 9,534 (30.6%) | 9.658 (31.0%) | -0.0093 | 16,081 (32.7%) | 16,255 (33.1%) | -0.003 |
| OCM - Dorsopathies: n (%) | 5,053 (28.0%) | 5,104 (28.3%) | -0.0067 | 7,003 (22.5%) | 7.086 (22.8%) | -0.0072 | 12,056 (24.5%) | 12,190 (24.8%) | -0.007 |
| OCM-Gout (acute/chronic); n (%)* | 121 (0.7%) | 143 (0.8%) | -0.0116 | 238 (0.8%) | 227 (0.7%) | 0.0116 | 359 (0.7%) | 370 (0.8%) | -0.012 |
| OCM-Hyperthyroidism ; n (%)* | 121 (0.7%) | 107 (0.6%) | 0.0124 | 145 (0.5%) | 142 (0.5%) | 0.0000 | 266 (0.5%) | 249 (0.5%) | 0.000 |
| OCM-Hypothyroidism; n (%)* | 1,760 (9.8%) | 1,783 (9.9%) | -0.0034 | 2,214 (7.1%) | 2,255 (7.2%) | -0.0039 | 3,974 (8.1%) | 4,038 (8.2%) | -0.004 |
| OCM-VTE; n (%)* | 333 (1.8%) | 337 (1.9%) | -0.0074 | 570 (1.8%) | 583 (1.9%) | -0.0074 | 903 (1.8%) | 920 (1.9%) | -0.007 |
| OCM-GERD; n (%) | 2,541 (14.1%) | 2,518 (14.0%) | 0.0029 | 2,368 (7.6%) | 2,363 (7.6%) | 0.0000 | 4,909 (10.0%) | 4,881 (9.9%) | 0.003 |
| OCM-Cancer; n (%) | 1,869 (10.4%) | 1,909 (10.6%) | -0.0065 | 2,579 (8.3%) | 2,626 (8.4%) | -0.0036 | 4,448 (9.1%) | 4,535 (9.2%) | -0.003 |
| OCM - Hypovolemia/volume depletion ; n (%)* OCM - Anemia ; n (%) | 383 (2.1%)<br>1,830 (10.2%) | 404 (2.2%)<br>1,853 (10.3%) | -0.0069<br>-0.0033 | 523 (1.7%)<br>2,414 (7.8%) | 558 (1.8%)<br>2,460 (7.9%) | -0.0076<br>-0.0037 | 906 (1.8%)<br>4,244 (8.6%) | 962 (2.0%)<br>4,313 (8.8%) | -0.015<br>-0.007 |
| OCM-Dementia:n(%)* | 1,830 (10.2%)<br>639 (3.5%) | 763 (4.2%) | -0.0364 | 751 (2.4%) | 916 (2.9%) | -0.0037 | 1,390 (2.8%) | 1,679 (3.4%) | -0.007 |
| OCM - Derression ; n (%) | 2,800 (15.5%) | 2,815 (15.6%) | -0.0028 | 2,980 (9.6%) | 2,938 (9.4%) | 0.0068 | 5,780 (11.8%) | 5,753 (11.7%) | 0.003 |
| Sum Supression ; in (vi) | 2,000 (13.370) | 2,013 (13.070) | | 2,550 (5.670) | 2,550 (5.476) | | 27. 22 (22.2.2) | 5,100 (2011) | |
| ORX - Metformin; n (%)* | 1,839 (10.2%) | 1,854 (10.3%) | -0.0033 | 2,684 (8.6%) | 2,719 (8.7%) | -0.0036 | 4,523 (9.2%) | 4,573 (9.3%) | -0.003 |
| ORX - 1st and 2nd Generation SUs ; n (%) | 896 (5.0%) | 922 (5.1%) | -0.0046 | 1,594 (5.1%) | 1,545 (5.0%) | 0.0046 | 2,490 (5.1%) | 2,467 (5.0%) | 0.005 |
| ORX - Insulins ; n (%) | 755 (4.2%) | 776 (4.3%) | -0.0050 | 1,328 (4.3%) | 1,333 (4.3%) | 0.0000 | 2,083 (4.2%) | 2,109 (4.3%) | -0.005 |
| ORX - Other antidiabetic medications use; n (%) | 683 (3.8%) | 662 (3.7%) | 0.0053 | 1,486 (4.8%) | 1,481 (4.8%) | 0.0000 | 2,169 (4.4%) | 2,143 (4.4%) | 0.000 |
| ORX - PPIs or H2RAs use; n (%)* | 4,194 (23.3%) | 4,378 (24.3%) | -0.0235 | 6,598 (21.2%) | 6,855 (22.0%) | -0.0194 | 10,792 (22.0%) | 11,233 (22.9%) | -0.022 |
| ORX - NSAIDs ; n (%)* ORX - Use of opioids ; n (%)* | 2,930 (16.3%)<br>6,320 (35.1%) | 3,002 (16.7%)<br>6,310 (35.0%) | -0.0108<br>0.0021 | 5,255 (16.9%)<br>11,650 (37.4%) | 5,441 (17.5%)<br>11,206 (36.0%) | -0.0159<br>0.0290 | 8,185 (16.7%)<br>17,970 (36.6%) | 8,443 (17.2%)<br>17,516 (35.6%) | -0.013<br>0.021 |
| ORX - Use of opioids ; n (%)* | 815 (4.5%) | 809 (4.5%) | 0.0021 | 1,220 (3.9%) | 1,219 (3.9%) | 0.0000 | 2,035 (4.1%) | 2,028 (4.1%) | 0.000 |
| ORX - Use of antidepressants : n (%) | 6,448 (35.8%) | 6,479 (36.0%) | -0.0042 | 10,791 (34.7%) | 10,840 (34.8%) | -0.0021 | 17,239 (35.1%) | 17,319 (35.2%) | -0.002 |
| ORX - Use of anxiolytics/hypnotics ; n (%) | 1,758 (9.8%) | 1,771 (9.8%) | 0.0000 | 3,350 (10.8%) | 3,360 (10.8%) | 0.0000 | 5,108 (10.4%) | 5,131 (10.4%) | 0.000 |
| ORX - Use of anticonvulsants ; n (%)* | 3,002 (16.7%) | 2,999 (16.6%) | 0.0027 | 4,192 (13.5%) | 4,186 (13.5%) | 0.0000 | 7,194 (14.6%) | 7,185 (14.6%) | 0.000 |
| ORX - Use of Benzodiazepines ; n (%)* | 3,043 (16.9%) | 2,933 (16.3%) | 0.0161 | 7,066 (22.7%) | 6,761 (21.7%) | 0.0241 | 10,109 (20.6%) | 9,694 (19.7%) | 0.022 |
| ORX - Use of dementia meds ; n (%)* | 451 (2.5%) | 528 (2.9%) | -0.0247 | 744 (2.4%) | 906 (2.9%) | -0.0311 | 1,195 (2.4%) | 1,434 (2.9%) | -0.031 |
| ORX - Use of antiparkinsonian meds ; n (%)* | 686 (3.8%) | 657 (3.6%) | 0.0106 | 1,028 (3.3%) | 1,055 (3.4%) | -0.0056 | 1,714 (3.5%) | 1,712 (3.5%) | 0.000 |
| ORX - Use of oral anticoagulants ; n (%)* | 879 (4.9%) | 891 (4.9%) | 0.0000 | 1,774 (5.7%) | 1,819 (5.8%) | -0.0043 | 2,653 (5.4%) | 2,710 (5.5%) | -0.004 |
| ORX - Use of antiplatelet agents ; n (%)* | 1,174 (6.5%) | 1,104 (6.1%) | 0.0165 | 3,085 (9.9%) | 2,922 (9.4%) | 0.0169 | 4,259 (8.7%) | 4,026 (8.2%) | 0.018 |
| LFS - Obesity; n (%) | 1,298 (7.2%) | 1,310 (7.3%) | -0.0039 | 1,289 (4.1%) | 1,290 (4.1%) | 0.0000 | 2,587 (5.3%) | 2,600 (5.3%) | 0.000 |
| · | | | | | | | 10,260 (20.9%) | 0.000/20.20/ | 0.015 |
| DET - Spirometry test only: n (%) | 3 100 (17 60/) | 3 038 /16 00/1 | 0.0212 | | | | | | |
| PFT - Spirometry test only; n (%) PFT - Spirometry test only (Count - 180 days to 31 days before CED) * | 3,180 (17.6%) | 3,028 (16.8%) | 0.0212 | 7,080 (22.7%) | 6,932 (22.3%) | 0.0096 | | 9,960 (20.3%) | |
| | 3,180 (17.6%)<br>0.18 (0.66)<br>0.00 [0.00, 0.00] | 3,028 (16.8%)<br>0.18 (0.65)<br>0.00 [0.00, 0.00] | 0.0212<br>0.0000<br>0.0000 | 7,080 (22.7%)<br>0.20 (0.64)<br>0.00 [0.00, 0.00] | 6,932 (22.3%)<br>0.22 (0.65)<br>0.00 [0.00, 0.00] | -0.0310<br>0.0000 | 0.19 (0.65)<br>0.00 (0.65) | 0.21 (0.65)<br>0.00 (0.65) | -0.031<br>0.000 |

| mean (sd) | 0.14 (0.56) | 0.11 (0.48) | 0.0575 | 0.17 (0.55) | 0.13 (0.47) | 0.0782 | 0.16 (0.55) | 0.12 (0.47) | 0.078 |
|---|---|---|---|---|---|---|---|---|---|
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.55) | 0.00 (0.47) | 0.000 |
| PFT - Lung volume, Diffuse capacity, pulmonary stress testing (any); n (%) | 1,987 (11.0%) | 1,910 (10.6%) | 0.0129 | 3,084 (9.9%) | 2,970 (9.5%) | 0.0135 | 5,071 (10.3%) | 4,880 (9.9%) | 0.013 |
| g in g | , | , | | γ , | , , , , , | | | | |
| HCU - Pulmonologist visit (180 to 1 day before CED); n (%) | 189 (1.0%) | 182 (1.0%) | 0.0000 | 5,646 (18.1%) | 5,482 (17.6%) | 0.0131 | 5,835 (11.9%) | 5,664 (11.5%) | 0.012 |
| HCU - Pulmonologist visit on CED; n (%) | 24 (0.1%) | 24 (0.1%) | 0.0000 | 949 (3.0%) | 932 (3.0%) | 0.0000 | 973 (2.0%) | 956 (1.9%) | 0.007 |
| HCU - Pulmonologist visit (Number of during CAP) * | ' ' | ` ' | | · · | ` ' | | | | |
| mean (sd) | 0.06 (0.94) | 0.07 (0.94) | -0.0106 | 0.75 (2.21) | 0.70 (2.11) | 0.0231 | 0.50 (1.85) | 0.47 (1.77) | 0.017 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (1.85) | 0.00 (1.77) | 0.000 |
| HCU - Number of Internal Medicine/Family Medicine Visits | | | | | | | | | |
| mean (sd) | 7.48 (11.28) | 7.62 (11.09) | -0.0125 | 6.14 (9.32) | 6.16 (9.74) | -0.0021 | 6.63 (10.08) | 6.70 (10.26) | -0.007 |
| median [IQR] | 4.00 [1.00, 10.00] | 4.00 [1.00, 10.00] | 0.0000 | 4.00 [1.00, 8.00] | 3.00 [1.00, 8.00] | 0.1049 | 4.00 (10.08) | 3.37 (10.26) | 0.062 |
| HCU - Number of Cardiologist visits | | | | | | | | | |
| mean (sd) | 0.86 (3.19) | 0.86 (2.82) | 0.0000 | 0.79 (2.82) | 0.79 (3.36) | 0.0000 | 0.82 (2.96) | 0.82 (3.17) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (2.96) | 0.00 (3.17) | 0.000 |
| HCU - Number of Emergency Department (ED) visits v3 | | | | | | | | | |
| mean (sd) | 0.46 (1.29) | 0.47 (1.25) | -0.0079 | 0.17 (1.12) | 0.16 (0.95) | 0.0096 | 0.28 (1.19) | 0.27 (1.07) | 0.009 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (1.19) | 0.00 (1.07) | 0.000 |
| HCU - Old hospitalization (-180 days to -31 days before CED); n (%) | 1,508 (8.4%) | 1,514 (8.4%) | 0.0000 | 4,137 (13.3%) | 4,095 (13.2%) | 0.0029 | 5,645 (11.5%) | 5,609 (11.4%) | 0.003 |
| HCU - Recent hospitalization (-30 days to CED date); n (%) | 166 (0.9%) | 166 (0.9%) | 0.0000 | 532 (1.7%) | 523 (1.7%) | 0.0000 | 698 (1.4%) | 689 (1.4%) | 0.000 |
| HCU - Number of hospitalizations during CAP | | | | | | | | | |
| mean (sd) | 0.11 (0.37) | 0.11 (0.37) | 0.0000 | 0.17 (0.43) | 0.16 (0.43) | 0.0233 | 0.15 (0.41) | 0.14 (0.41) | 0.024 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.41) | 0.00 (0.41) | 0.000 |
| HCU - Blood eosinophilia or Serum IgE test order; n (%)* | 85 (0.5%) | 93 (0.5%) | 0.0000 | 113 (0.4%) | 136 (0.4%) | 0.0000 | 198 (0.4%) | 229 (0.5%) | -0.015 |
| HCU - Pneumococcal vaccine; n (%) | 2,119 (11.8%) | 2,112 (11.7%) | 0.0031 | 1,615 (5.2%) | 1,601 (5.1%) | 0.0045 | 3,734 (7.6%) | 3,713 (7.6%) | 0.000 |
| HCU - Flu vaccine ; n (%) | 3,385 (18.8%) | 3,370 (18.7%) | 0.0026 | 3,684 (11.8%) | 3,659 (11.8%) | 0.0000 | 7,069 (14.4%) | 7,029 (14.3%) | 0.003 |
| HCU - Bone mineral density ; n (%) | 795 (4.4%) | 788 (4.4%) | 0.0000 | 931 (3.0%) | 953 (3.1%) | -0.0058 | 1,726 (3.5%) | 1,741 (3.5%) | 0.000 |
| HCU - Pap smear; n (%) | 711 (3.9%) | 707 (3.9%) | 0.0000 | 1,429 (4.6%) | 1,419 (4.6%) | 0.0000 | 2,140 (4.4%) | 2,126 (4.3%) | 0.005 |
| HCU - Mammogram ; n (%) | 2,274 (12.6%) | 2,273 (12.6%) | 0.0000 | 3,319 (10.7%) | 3,340 (10.7%) | 0.0000 | 5,593 (11.4%) | 5,613 (11.4%) | 0.000 |
| HCU - Prostate exam for DRE; n (%) | 542 (3.0%) | 545 (3.0%) | 0.0000 | 517 (1.7%) | 509 (1.6%) | 0.0079 | 1,059 (2.2%) | 1,054 (2.1%) | 0.007 |
| HCU - Number of Echocardiogram * | | | | | | | | | |
| mean (sd) | 0.20 (1.27) | 0.19 (1.21) | 0.0081 | 0.23 (0.80) | 0.23 (0.84) | 0.0000 | 0.22 (1.00) | 0.22 (0.99) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (1.00) | 0.00 (0.99) | 0.000 |
| HCU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy ; n (%) | 816 (4.5%) | 808 (4.5%) | 0.0000 | 1,609 (5.2%) | 1,634 (5.3%) | -0.0045 | 2,425 (4.9%) | 2,442 (5.0%) | -0.005 |
| HCU - Number of Distinct Medication Prescriptions (not generalized to generics) | | | | | | | | | |
| mean (sd) | 20.27 (17.04) | 20.34 (16.67) | -0.0042 | 19.34 (15.01) | 19.39 (15.01) | -0.0033 | 19.68 (15.78) | 19.74 (15.64) | -0.004 |
| median [IQR] | 16.00 [8.00, 27.00] | 16.00 [9.00, 27.00] | 0.0000 | 16.00 [9.00, 26.00] | 16.00 [9.00, 26.00] | 0.0000 | 16.00 (15.78) | 16.00 (15.64) | 0.000 |
| SES - Copay for pharmacy cost (charges in U.S. \$) | | | | | | | | | |
| mean (sd) | 32.00 (38.05) | 31.87 (35.15) | 0.0035 | 25.66 (26.01) | 25.75 (26.16) | -0.0035 | 27.98 (30.97) | 27.99 (29.77) | 0.000 |
| median [IQR] | 23.60 [10.60, 40.25] | 24.23 [10.04, 41.52] | -0.0172 | 20.26 [10.00, 34.37] | 20.61 [9.80, 34.59] | -0.0134 | 21.48 (30.97) | 21.94 (29.77) | -0.015 |
| SES - Business type | | | | | | | | | |
| Commercial; n (%) | 5,963 (33.1%) | 5,735 (31.8%) | 0.0278 | | | | 5,963 (33.1%) | 5,735 (31.8%) | 0.028 |
| Medicare; n (%) | 12,054 (66.9%) | 12,282 (68.2%) | -0.0278 | | | $\perp$ | 12,054 (66.9%) | 12,282 (68.2%) | -0.028 |
| SES - Low income indicator ; n (%) | 3,483 (19.3%) | 3,604 (20.0%) | -0.0176 | | | $\perp$ | 3,483 (19.3%) | 3,604 (20.0%) | -0.018 |
| SES - Insurance Plan type | | | | | | | | | |
| Comprehensive; n (%) | | | | 9,074 (29.2%) | 9,146 (29.4%) | -0.0044 | 9,074 (29.2%) | 9,146 (29.4%) | -0.004 |
| HMO; n (%) | | | | 3,810 (12.2%) | 3,763 (12.1%) | 0.0031 | 3,810 (12.2%) | 3,763 (12.1%) | 0.003 |
| PPO; n (%) | | | | 14,372 (46.2%) | 14,423 (46.3%) | -0.0020 | 14,372 (46.2%) | 14,423 (46.3%) | -0.002 |
| Others; n (%) | | | | 3,866 (12.4%) | 3,790 (12.2%) | 0.0061 | 3,866 (12.4%) | 3,790 (12.2%) | 0.006 |

<sup>\*</sup> Not included in PS model